CLINICAL TRIAL: NCT01144663
Title: Immunogenicity and Safety of GSK Biologicals' Meningococcal Vaccine (GSK 134612) When Co-administered With a Pneumococcal Conjugate Vaccine and Infanrix Hexa™ in Healthy Infants
Brief Title: Immunogenicity and Safety of Meningococcal Vaccine GSK 134612 Co-administered With Pneumococcal and DTPa-HBV-IPV/Hib Vaccines
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 113369; 2009-016841-24 (EudraCT Number)
Record Dates: First submitted 2010-06-03; First posted 2010-06-15 (Estimated); Results first posted 2019-02-01 (Actual); Last update posted 2020-12-31 (Actual); Status verified 2020-12

CONDITIONS: Infections, Meningococcal; Meningococcal Vaccines
Keywords: Infants; conjugate vaccine; immunogenicity; meningococcal vaccine; non-inferiority; co-administration
MeSH Terms: conditions — Meningococcal Infections | interventions — diphtheria-tetanus-acellular pertussis-inactivated poliovirus-Haemophilus influenzae b conjugate-hepatitis B vaccine; PHiD-CV vaccine

ARMS (4):
- Nimenrix 3 Group (Experimental): Healthy male or female subjects aged between and including, 6 and 12 weeks of age, intramuscularly received 3 primary doses of Nimenrix™ vaccine at 2, 3 and 4 months of age, followed by a booster dose of Nimenrix™ vaccine at 12 months of age. Subjects were also administered intramuscular injections of Infanrix™ hexa and Synflorix™ vaccines at 2, 3, 4 and 12 months of age.
  Interventions: Biological: Nimenrix™; Biological: Infanrix™ hexa; Biological: Synflorix™
- Nimenrix 2 Group (Experimental): Healthy male or female subjects aged between and including, 6 and 12 weeks of age, intramuscularly received 2 primary doses of Nimenrix™ vaccine at 2 and 4 months of age, followed by a booster dose of Nimenrix™ vaccine at 12 months of age. Subjects were also administered intramuscular injections of Infanrix™ hexa and Synflorix™ vaccines at 2, 4 and 12 months of age.
  Interventions: Biological: Nimenrix™; Biological: Infanrix™ hexa; Biological: Synflorix™
- Menjugate Group (Active Comparator): Healthy male or female subjects aged between and including, 6 and 12 weeks of age, intramuscularly received 2 primary doses of Menjugate® vaccine at 2 and 4 months of age, followed by a booster dose of Menjugate® vaccine at 12 months of age. Subjects were also administered intramuscular injections of Infanrix™ hexa and Synflorix™ vaccines at 2, 4 and 12 months of age.
  Interventions: Biological: Menjugate®; Biological: Infanrix™ hexa; Biological: Synflorix™
- NeisVac-C Group (Active Comparator): Healthy male or female subjects aged between and including, 6 and 12 weeks of age, intramuscularly received 2 primary doses of NeisVac-C™ vaccine at 2 and 4 months of age, followed by a booster dose of NeisVac-C™ vaccine at 12 months of age. Subjects were also administered intramuscular injections of Infanrix™ hexa and Synflorix™ vaccines at 2, 4 and 12 months of age.
  Interventions: Biological: NeisVac-CTM; Biological: Infanrix™ hexa; Biological: Synflorix™

INTERVENTIONS:
Biological: Nimenrix™ — 4- or 3-dose intramuscular injection
  Arms: Nimenrix 2 Group; Nimenrix 3 Group
Biological: Menjugate® — 3-dose intramuscular injection
  Arms: Menjugate Group
Biological: NeisVac-CTM — 3-dose intramuscular injection
  Arms: NeisVac-C Group
Biological: Infanrix™ hexa — 4-dose intramuscular injection
  Other Names: Infanrix hexa™
Biological: Synflorix™ — 4-dose intramuscular injection

SUMMARY:
The purpose of this study is to evaluate immunogenicity and safety of meningococcal conjugate vaccine GSK134612 compared to the licensed vaccines MenC-CRM197 and MenC-TT in infants of 2 months of age. Pneumococcal conjugate vaccine and DTPa-HBV-IPV/Hib vaccines will be co-administered.

DETAILED DESCRIPTION:
The study consists of a primary vaccination phase and a booster vaccination phase. The Protocol Posting has been updated due to protocol amendment 2.

ELIGIBILITY:
Inclusion Criteria:

All subjects must satisfy ALL the following criteria at study entry:

* Subjects who the investigator believes that their parent(s)/Legally Acceptable Representative(s) (LAR) can and will comply with the requirements of the protocol (e.g. completion of the diary cards, return for follow-up visit).
* A male or female between, and including, 6 and 12 weeks (42-90 days) of age at the time of the first vaccination.
* Written informed consent obtained from the parent(s) or guardian of the subject.
* Free of obvious health problems as established by medical history and clinical examination before entering into the study.
* Born after a gestation period of at least 36 weeks.

Exclusion Criteria:

* Child in care.
* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine(s) within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Extended administration (defined as more than 14 days in total) of immunosuppressants or other immune-modifying drugs since birth. For corticosteroids, this will mean prednisone >= 0.5 mg/kg/day, or equivalent. Inhaled and topical steroids are allowed.
* Planned administration/ administration of a vaccine not foreseen by the study protocol during the period starting 30 days before the first dose of vaccine(s) until 30 days after the last dose of vaccine(s) (i.e. booster dose), with the exception of rotavirus vaccine which can be administered at any time during the study, according to the national immunisation recommendations. MMR(V) vaccine, if recommended in national immunisation programs, can be given after the last blood sampling time point i.e. after Visit 6. Seasonal or pandemic influenza vaccine can be given at any time during the study, and according to the Summary of Product Characteristics and national recommendations.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product (pharmaceutical product or device).
* Previous vaccination against diphtheria, tetanus, pertussis, polio, hepatitis B, Haemophilus influenzae type b, Streptococcus pneumoniae, Neisseria meningitidis serogroups A, C, W-135 or Y with the exception of vaccines where the first dose may be given within the first two weeks of life according to the national recommendations (for example hepatitis B and BCG).
* History of, or intercurrent, diphtheria, tetanus, pertussis, polio, hepatitis B, Haemophilus influenzae type b disease, pneumococcal and/or meningococcal disease.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination (no laboratory testing required).
* Family history of congenital or hereditary immunodeficiency.
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the vaccine(s).
* Major congenital defects or serious chronic illness.
* History of any neurologic disorders or seizures (history of a single, simple febrile seizure is permitted).
* Acute disease and/or fever at the time of enrolment. (Fever is defined as temperature ≥ 37.5°C (99.5°F) on oral, axillary or tympanic setting, or ≥ 38.0°C (100.4°F) on rectal setting).

(Subjects with a minor illness (such as mild diarrhoea, mild upper respiratory infection) without fever may, be enrolled at the discretion of the investigator).

- Administration of immunoglobulins and/ or any blood products since birth or planned administration during the study period.

Ages: 6 Weeks to 12 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2095 (Actual)
Dates: Start 2010-07-01 (Actual); Primary Completion 2012-06-22 (Actual); Study Completion 2013-09-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (40):
- Estonia (3):
  - GSK Investigational Site, Haabneeme
  - GSK Investigational Site, Tallinn
  - GSK Investigational Site, Tartu
- Germany (26):
  - GSK Investigational Site, Kehl, Baden-Wurttemberg
  - GSK Investigational Site, Schwäbisch Hall, Baden-Wurttemberg
  - GSK Investigational Site, Berchtesgaden, Bavaria
  - GSK Investigational Site, Bindlach, Bavaria
  - GSK Investigational Site, Gilching, Bavaria
  - GSK Investigational Site, Kirchheim, Bavaria
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Weilheim, Bavaria
  - GSK Investigational Site, Baunatal-Grossenritte, Hesse
  - GSK Investigational Site, Eschwege, Hesse
  - GSK Investigational Site, Vellmar, Hesse
  - GSK Investigational Site, Detmold, North Rhine-Westphalia
  - GSK Investigational Site, Kleve-Materborn, North Rhine-Westphalia
  - GSK Investigational Site, Porta Westfalica, North Rhine-Westphalia
  - GSK Investigational Site, Solingen, North Rhine-Westphalia
  - GSK Investigational Site, Frankenthal, Rhineland-Palatinate
  - GSK Investigational Site, Mainz, Rhineland-Palatinate
  - GSK Investigational Site, Trier, Rhineland-Palatinate
  - GSK Investigational Site, Worms, Rhineland-Palatinate
  - GSK Investigational Site, Leipzig, Saxony
  - GSK Investigational Site, Wurzen, Saxony
  - GSK Investigational Site, Wanzleben, Saxony-Anhalt
  - GSK Investigational Site, Weißenfels, Saxony-Anhalt
  - GSK Investigational Site, Flensburg, Schleswig-Holstein
  - GSK Investigational Site, Bad Lobenstein, Thuringia
  - GSK Investigational Site, Berlin
- Spain (11):
  - GSK Investigational Site, Almería
  - GSK Investigational Site, Antequera/Málaga
  - GSK Investigational Site, Badalona
  - GSK Investigational Site, Blanes (Girona)
  - GSK Investigational Site, Burgos
  - GSK Investigational Site, Ciudad Real
  - GSK Investigational Site, Manlleu
  - GSK Investigational Site, Seville
  - GSK Investigational Site, Valencia
  - GSK Investigational Site, Valladolid
  - GSK Investigational Site, Vic

REFERENCES:
- [Background] Merino Arribas JM, Carmona Martinez A, Horn M, Perez Porcuna XM, Otero Reigada MD, Mares Bermudez J, Centeno Malfaz F, Miranda M, Mendez M, Garcia Cabezas MA, Wittermann C, Bleckmann G, Fischbach T, Kolhe D, van der Wielen M, Baine Y. Safety and Immunogenicity of the Quadrivalent Meningococcal Serogroups A, C, W and Y Tetanus Toxoid Conjugate Vaccine Coadministered With Routine Childhood Vaccines in European Infants: An Open, Randomized Trial. Pediatr Infect Dis J. 2017 Apr;36(4):e98-e107. doi: 10.1097/INF.0000000000001484. PMID 28002359
- [Background] Merino Arribas JM, Carmona Martinez A, Horn M, Perez Porcuna XM, Otero Reigada MDC, Mares Bermudez J, Centeno Malfaz F, Miranda M, Mendez M, Garcia Cabezas MA, Christoph W, Bleckmann G, Fischbach T, Kolhe D, Van der Wielen M, Baine Y. Immunogenicity and Reactogenicity of DTPa-HBV-IPV/Hib and PHiD-CV When Coadministered With MenACWY-TT in Infants: Results of an Open, Randomized Trial. Pediatr Infect Dis J. 2018 Jul;37(7):704-714. doi: 10.1097/INF.0000000000002061. PMID 29620722

RESULTS

PARTICIPANT FLOW:
Period: Primary Vaccination Phase
Arm/Group | Nimenrix 3 Group | Nimenrix 2 Group | Menjugate Group | NeisVac-C Group
Started | 528 | 524 | 516 | 527
Completed | 508 | 517 | 508 | 509
Not Completed | 20 | 7 | 8 | 18
Not completed — Serious adverse event, fatal | 2 | 0 | 1 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 1
Not completed — Protocol Violation | 2 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 9 | 5 | 3 | 10
Not completed — Migrated/moved from study area | 4 | 1 | 2 | 3
Not completed — Lost to Follow-up | 2 | 0 | 1 | 2
Not completed — Other | 0 | 1 | 0 | 2
Period: Booster Vaccination Phase
Arm/Group | Nimenrix 3 Group | Nimenrix 2 Group | Menjugate Group | NeisVac-C Group
Started | 497 | 511 | 503 | 506
Completed | 494 | 509 | 498 | 505
Not Completed | 3 | 2 | 5 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 1
Not completed — Migrated/moved from study area | 1 | 1 | 1 | 0
Not completed — Lost to Follow-up | 2 | 1 | 3 | 0
Period: Extended Safety Follow-Up (ESFU)
Arm/Group | Nimenrix 3 Group | Nimenrix 2 Group | Menjugate Group | NeisVac-C Group
Started | 497 | 511 | 503 | 506
Completed | 492 | 502 | 496 | 505
Not Completed | 5 | 9 | 7 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 1
Not completed — Migrated/moved from study area | 1 | 3 | 1 | 0
Not completed — Lost to Follow-up | 4 | 6 | 5 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nimenrix 3 Group | Nimenrix 2 Group | Menjugate Group | NeisVac-C Group | Total
Number analyzed (Participants) | 528 | 524 | 516 | 527 | 2095
Age, Continuous [Mean (Standard Deviation); unit: Weeks] | 8.7 (1.54) | 8.6 (1.52) | 8.7 (1.53) | 8.6 (1.49) | 8.65 (1.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 255 | 273 | 264 | 251 | 1043
  Male | 273 | 251 | 252 | 276 | 1052
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Geographic ancestry: African heritage/African American | 5 | 4 | 6 | 1 | 16
  Geographic ancestry: American Indian or Alaskan Native | 1 | 4 | 4 | 2 | 11
  Geographic ancestry: Asian-Central/South Asian heritage | 1 | 1 | 0 | 0 | 2
  Geographic ancestry: Asian-East Asian heritage | 0 | 1 | 1 | 1 | 3
  Geographic ancestry: Asian-South East Asian heritage | 1 | 0 | 0 | 0 | 1
  Geographic ancestry: Native Hawaiian or other Pacific Islander | 0 | 0 | 1 | 0 | 1
  Geographic ancestry: White-Arabic/North African heritage | 12 | 8 | 10 | 21 | 51
  Geographic ancestry: White-Caucasian/European heritage | 500 | 497 | 486 | 495 | 1978
  Geographic ancestry: Not specified | 8 | 9 | 8 | 7 | 32

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With Serum Bactericidal Assay Using Baby Rabbit Complement Against Meningococcal Serogroups A, W-135 and Y (rSBA-MenA, rSBA-MenW-135 and rSBA-Y) Antibody Titers Greater Than or Equal to (≥) the Cut-off Value.
Description: The cut-off value for the rSBA-MenA, rSBA-MenW-135 and rSBA-Y titers was greater than or equal to (≥) 1:8.
  Indication of the immunogenicity of the 2-dose and 3-dose schedules: the lower limit of the two-sided exact 95% CI for the percentage of subjects with post-primary vaccination rSBA antibody titre ≥ 1:8 is greater than or equal to the pre-defined clinical limit of 80%.
Time Frame: One month after the final primary vaccination at Month 3
Population: The analysis was performed on the Primary According-to-Protocol (ATP) cohort for immunogenicity, including all subjects who complied with the protocol, who were administered a vaccine containing rSBA-MenA, rSBA-MenW-135 and rSBA-Y components (i.e. only Group Nimenrix 3 and Nimenrix 2) and with available data for the considered assay and time point.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Nimenrix 3 Group | Nimenrix 2 Group
Number analyzed (Participants) | 462 | 456
Percentage of Participants
  rSBA-MenA | 99.4 [98.1 to 99.9] | 97.4 [95.4 to 98.6]
  rSBA-MenW-135: number analyzed (Participants) | 461 | 455
  rSBA-MenW-135 | 99.1 [97.8 to 99.8] | 99.1 [97.8 to 99.8]
  rSBA-MenY: number analyzed (Participants) | 461 | 456
  rSBA-MenY | 93.1 [90.3 to 95.2] | 98.2 [96.6 to 99.2]

2. Primary Outcome: Number of Subjects With rSBA-MenC Antibody Titers ≥ the Cut-off Value
Description: The cut-off value for rSBA-MenC titers was ≥ 1:8.
Time Frame: One month after the final primary vaccination at Month 3
Population: The analysis was performed on the Primary ATP cohort for immunogenicity, which included all evaluable subjects who complied with the vaccination schedule for Visit 1, 2 and 3 (Day 0 to Month 2)and with the blood sample schedule for Visit 4 (Month 3).
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix 3 Group | Nimenrix 2 Group | Menjugate Group | NeisVac-C Group
Number analyzed (Participants) | 461 | 456 | 455 | 457
Participants | 459 | 450 | 453 | 457
Statistical Analysis 1: Comparison: Nimenrix 3 Group vs Menjugate Group; To demonstrate the non-inferiority of the Nimenrix 3 Group compared to the Menjugate Group, two-sided standardized asymptotic 95% CI (confidence interval) for the groups difference [Nimenrix 3 Group minus Menjugate Group] in the percentages of subjects with bactericidal vaccine response to MenC was computed; Test type: Non-Inferiority — Indication of non-inferiority of Nimenrix 3 Group compared to Menjugate Group is a lower limit of the 95% CI of the group difference greater than or equal to the predefined clinical limits of -5%; Difference in percentage = 0.01, 95% CI 2-sided [-1.17 to 1.2]
Statistical Analysis 2: Comparison: Nimenrix 3 Group vs NeisVac-C Group; To demonstrate the non-inferiority of the Nimenrix 3 Group compared to the NeisVac-C Group, two-sided standardized asymptotic 95% CI for the groups difference [Nimenrix 3 Group minus NeisVac-C Group] in the percentages of subjects with bactericidal vaccine response to MenC was computed; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; Difference in percenttage = -0.43, 95% CI 2-sided [-1.57 to 0.4]
Statistical Analysis 3: Comparison: Nimenrix 2 Group vs Menjugate Group; To demonstrate the non-inferiority of the Nimenrix 2 Group compared to Menjugate Group, two-sided standardized asymptotic 95% CI for the groups difference [Nimenrix 2 Group minus Menjugate Group] in the percentages of subjects with bactericidal vaccine response to MenC was computed; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; Difference in percentage = -0.88, 95% CI 2-sided [-2.45 to 0.43]
Statistical Analysis 4: Comparison: Nimenrix 2 Group vs NeisVac-C Group; To demonstrate the non-inferiority of the Nimenrix 2 Group compared to NeisVac-C Group, two-sided standardized asymptotic 95% CI for the groups difference [Nimenrix 2 Group minus NeisVac-C Group] in the percentages of subjects with bactericidal vaccine response to MenC was computed; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; Difference in percentage = -1.32, 95% CI 2-sided [-2.84 to -0.48]

3. Secondary Outcome: Number of Subjects With rSBA-MenA, rSBA-MenC, rSBA-MenW-135 and rSBA-MenY Titers Above Cut-off Values
Description: The cut-off values for rSBA-Men antibody titers were greater than or equal to (≥) 1:8 and ≥ 1:128 at pre-vaccination
Time Frame: Pre-primary vaccination at Month 0
Population: The analysis was performed on the Primary ATP cohort for immunogenicity, which included all evaluable subjects who complied with the vaccination schedule for a randomized subset of 50% subjects for each of the 4 serogroups in the investigational groups, and in a randomized subset of 50% and 25% subjects for MenC, MenA, MenW, MenY in control groups.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix 3 Group | Nimenrix 2 Group | Menjugate Group | NeisVac-C Group
Number analyzed (Participants) | 223 | 220 | 207 | 220
Participants
  rSBA-MenA ≥ 1:8: number analyzed (Participants) | 223 | 219 | 97 | 110
  rSBA-MenA ≥ 1:8 | 2 | 4 | 2 | 2
  rSBA-MenA ≥ 1:128: number analyzed (Participants) | 223 | 219 | 97 | 110
  rSBA-MenA ≥ 1:128 | 1 | 0 | 0 | 0
  rSBA-MenC ≥ 1:8 | 12 | 10 | 15 | 14
  rSBA-MenC ≥ 1:128 | 2 | 1 | 6 | 5
  rSBA-MenW-135 ≥ 1:8: number analyzed (Participants) | 215 | 217 | 110 | 107
  rSBA-MenW-135 ≥ 1:8 | 8 | 12 | 5 | 3
  rSBA-MenW-135 ≥ 1:128: number analyzed (Participants) | 215 | 217 | 110 | 107
  rSBA-MenW-135 ≥ 1:128 | 0 | 1 | 1 | 1
  rSBA-MenY ≥ 1:8: number analyzed (Participants) | 215 | 219 | 111 | 107
  rSBA-MenY ≥ 1:8 | 6 | 6 | 8 | 3
  rSBA-MenY ≥ 1:128: number analyzed (Participants) | 215 | 219 | 111 | 107
  rSBA-MenY ≥ 1:128 | 0 | 3 | 1 | 1

4. Secondary Outcome: rSBA-MenA, rSBA-MenC, rSBA-MenW-135 and rSBA-MenY Antibody Titers
Description: Antibody titers were presented as geometric mean titers (GMTs).
Time Frame: Pre-primary vaccination at Month 0
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Nimenrix 3 Group | Nimenrix 2 Group | Menjugate Group | NeisVac-C Group
Number analyzed (Participants) | 223 | 220 | 207 | 220
Titers
  rSBA-MenA: number analyzed (Participants) | 223 | 219 | 97 | 110
  rSBA-MenA | 4.1 [4 to 4.2] | 4.1 [4 to 4.2] | 4.1 [4 to 4.3] | 4.1 [3.9 to 4.3]
  rSBA-MenC | 4.4 [4.1 to 4.8] | 4.3 [4.1 to 4.5] | 4.9 [4.4 to 5.5] | 4.7 [4.3 to 5.2]
  rSBA-MenW-135: number analyzed (Participants) | 215 | 217 | 110 | 107
  rSBA-MenW-135 | 4.3 [4.1 to 4.5] | 4.4 [4.1 to 4.6] | 4.3 [3.9 to 4.8] | 4.3 [3.9 to 4.7]
  rSBA-MenY: number analyzed (Participants) | 215 | 219 | 111 | 107
  rSBA-MenY | 4.2 [4 to 4.4] | 4.2 [4 to 4.5] | 4.7 [4.2 to 5.2] | 4.2 [3.9 to 4.6]

5. Secondary Outcome: Number of Subjects With rSBA-MenA, rSBA-MenC, rSBA-MenW-135, rSBA-MenY Antibody Titers Above the Cut-off Values
Description: The cut-off values for the rSBA-Men antibody titers were greater than or equal to (≥) 1:8 and ≥ 1:128.
Time Frame: Pre-Booster dose at Month 10 and one month post-Booster dose at Month 11
Population: The analysis was performed on the Booster ATP cohort for immunogenicity, which included all evaluable subjects who complied with the vaccination schedule for Visit 5 (Month 10) and with blood sample schedule for Visit 6 (Month 11).
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix 3 Group | Nimenrix 2 Group | Menjugate Group | NeisVac-C Group
Number analyzed (Participants) | 441 | 463 | 446 | 461
Participants
  rSBA-MenA ≥ 1:8, Month 10: number analyzed (Participants) | 438 | 455 | 436 | 453
  rSBA-MenA ≥ 1:8, Month 10 | 300 | 279 | 26 | 23
  rSBA-MenA ≥ 1:128, Month 10: number analyzed (Participants) | 438 | 455 | 436 | 453
  rSBA-MenA ≥ 1:128, Month 10 | 107 | 99 | 11 | 3
  rSBA-MenA ≥ 1:8, Month 11: number analyzed (Participants) | 439 | 462 | 446 | 458
  rSBA-MenA ≥ 1:8, Month 11 | 437 | 460 | 21 | 19
  rSBA-MenA ≥ 1:128, Month 11: number analyzed (Participants) | 439 | 462 | 446 | 458
  rSBA-MenA ≥ 1:128, Month 11 | 433 | 456 | 8 | 12
  rSBA-MenC ≥ 1:8, Month 10: number analyzed (Participants) | 441 | 459 | 441 | 451
  rSBA-MenC ≥ 1:8, Month 10 | 324 | 348 | 229 | 356
  rSBA-MenC ≥ 1:128, Month 10: number analyzed (Participants) | 441 | 459 | 441 | 451
  rSBA-MenC ≥ 1:128, Month 10 | 108 | 183 | 79 | 195
  rSBA-MenC ≥ 1:8, Month 11: number analyzed (Participants) | 439 | 463 | 446 | 459
  rSBA-MenC ≥ 1:8, Month 11 | 437 | 462 | 439 | 459
  rSBA-MenC ≥ 1:128, Month 11: number analyzed (Participants) | 439 | 463 | 446 | 459
  rSBA-MenC ≥ 1:128, Month 11 | 432 | 454 | 426 | 457
  rSBA-MenW-135 ≥ 1:8, Month 10: number analyzed (Participants) | 441 | 459 | 440 | 453
  rSBA-MenW-135 ≥ 1:8, Month 10 | 372 | 417 | 18 | 27
  rSBA-MenW-135 ≥ 1:128, Month 10: number analyzed (Participants) | 441 | 459 | 440 | 453
  rSBA-MenW-135 ≥ 1:128, Month 10 | 221 | 254 | 16 | 22
  rSBA-MenW-135 ≥ 1:8, Month 11: number analyzed (Participants) | 437 | 462 | 445 | 459
  rSBA-MenW-135 ≥ 1:8, Month 11 | 433 | 461 | 34 | 37
  rSBA-MenW-135 ≥ 1:128, Month 11: number analyzed (Participants) | 437 | 462 | 445 | 459
  rSBA-MenW-135 ≥ 1:128, Month 11 | 430 | 457 | 31 | 31
  rSBA-MenY ≥ 1:8, Month 10: number analyzed (Participants) | 441 | 459 | 440 | 451
  rSBA-MenY ≥ 1:8, Month 10 | 364 | 383 | 54 | 47
  rSBA-MenY ≥ 1:128, Month 10: number analyzed (Participants) | 441 | 459 | 440 | 451
  rSBA-MenY ≥ 1:128, Month 10 | 126 | 168 | 41 | 37
  rSBA-MenY ≥ 1:8, Month 11: number analyzed (Participants) | 439 | 462 | 445 | 461
  rSBA-MenY ≥ 1:8, Month 11 | 436 | 459 | 45 | 40
  rSBA-MenY ≥ 1:128, Month 11: number analyzed (Participants) | 439 | 462 | 445 | 461
  rSBA-MenY ≥ 1:128, Month 11 | 419 | 445 | 37 | 34

6. Secondary Outcome: rSBA-MenA, rSBA-MenC, rSBA-MenW-135 and rSBA-MenY Antibody Titers
Description: Antibody titers were presented as geometric mean titers (GMTs).
Time Frame: Pre-Booster dose at Month 10 and one month post-Booster dose at Month 11
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Nimenrix 3 Group | Nimenrix 2 Group | Menjugate Group | NeisVac-C Group
Number analyzed (Participants) | 441 | 463 | 446 | 461
Titers
  rSBA-MenA, Month 10: number analyzed (Participants) | 438 | 455 | 436 | 453
  rSBA-MenA, Month 10 | 22.9 [19.8 to 26.5] | 19.5 [16.8 to 22.6] | 4.7 [4.3 to 5.0] | 4.4 [4.2 to 4.6]
  rSBA-MenA, Month 11: number analyzed (Participants) | 439 | 462 | 446 | 458
  rSBA-MenA, Month 11 | 1417.6 [1281.4 to 1568.3] | 1561.0 [1412.3 to 1725.3] | 4.6 [4.3 to 4.9] | 4.7 [4.3 to 5.0]
  rSBA-MenC, Month 10: number analyzed (Participants) | 441 | 459 | 441 | 451
  rSBA-MenC, Month 10 | 25.7 [22.3 to 29.6] | 43.7 [37.4 to 51.1] | 16.0 [13.8 to 18.5] | 49.3 [42.1 to 57.7]
  rSBA-MenC, Month 11: number analyzed (Participants) | 439 | 463 | 446 | 459
  rSBA-MenC, Month 11 | 1154.6 [1034.1 to 1289.0] | 1177.0 [1059.1 to 1308.0] | 1051.4 [919.6 to 1202.1] | 1960.2 [1776.4 to 2163.1]
  rSBA-MenW-135, Month 10: number analyzed (Participants) | 441 | 459 | 440 | 453
  rSBA-MenW-135, Month 10 | 68.7 [58.3 to 81.0] | 97.7 [83.3 to 114.5] | 4.7 [4.4 to 5.1] | 5.0 [4.6 to 5.5]
  rSBA-MenW-135, Month 11: number analyzed (Participants) | 437 | 462 | 445 | 459
  rSBA-MenW-135, Month 11 | 1955.9 [1729.6 to 2211.9] | 2777.2 [2485.1 to 3103.6] | 5.5 [5.0 to 6.1] | 5.6 [5.0 to 6.2]
  rSBA-MenY, Month 10: number analyzed (Participants) | 441 | 459 | 440 | 451
  rSBA-MenY, Month 10 | 35.4 [30.6 to 41.0] | 47.0 [40.3 to 54.7] | 6.5 [5.7 to 7.4] | 6.0 [5.4 to 6.8]
  rSBA-MenY, Month 11: number analyzed (Participants) | 439 | 462 | 445 | 461
  rSBA-MenY, Month 11 | 630.6 [564.1 to 705.1] | 881.3 [787.5 to 986.4] | 6.1 [5.4 to 6.8] | 5.8 [5.2 to 6.6]

7. Secondary Outcome: Number of Subjects With Serum Bactericidal Assay Using Human Complement Against Meningococcal Serogroups (hSBA-MenA, hSBA-MenC, hSBA-MenW-135 and hSBA-MenY) Antibody Titers Above the Cut-off Values
Description: The cut-off values for hSBA antibody titers were greater than or equal to (≥) 1:4 and ≥ 1:8.
Time Frame: Pre-primary vaccination at Month 0 and one month after final primary vaccination at Month 3
Population: The analysis was performed on the Primary ATP cohort for immunogenicity, which included all the evaluable subjects who used hSBA complement and who complied with the vaccination schedule for Visit 1, 2 and 3 (Day 0 to Month 2) and with the blood sample schedule for Visit 4 (Month 3).
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix 3 Group | Nimenrix 2 Group | Menjugate Group | NeisVac-C Group
Number analyzed (Participants) | 214 | 218 | 205 | 226
Participants
  hSBA-MenA ≥ 1:4, Month 0: number analyzed (Participants) | 164 | 166 | 161 | 166
  hSBA-MenA ≥ 1:4, Month 0 | 34 | 31 | 41 | 34
  hSBA-MenA ≥ 1:8, Month 0: number analyzed (Participants) | 164 | 166 | 161 | 166
  hSBA-MenA ≥ 1:8, Month 0 | 28 | 19 | 27 | 27
  hSBA-MenA ≥ 1:4, Month 3: number analyzed (Participants) | 200 | 202 | 172 | 205
  hSBA-MenA ≥ 1:4, Month 3 | 197 | 195 | 21 | 18
  hSBA-MenA ≥ 1:8, Month 3: number analyzed (Participants) | 200 | 202 | 172 | 205
  hSBA-MenA ≥ 1:8, Month 3 | 196 | 195 | 15 | 14
  hSBA-MenC ≥ 1:4, Month 0: number analyzed (Participants) | 181 | 178 | 168 | 185
  hSBA-MenC ≥ 1:4, Month 0 | 43 | 35 | 50 | 44
  hSBA-MenC ≥ 1:8, Month 0: number analyzed (Participants) | 181 | 178 | 168 | 185
  hSBA-MenC ≥ 1:8, Month 0 | 43 | 35 | 49 | 42
  hSBA-MenC ≥ 1:4, Month 3: number analyzed (Participants) | 214 | 218 | 202 | 226
  hSBA-MenC ≥ 1:4, Month 3 | 213 | 215 | 202 | 226
  hSBA-MenC ≥ 1:8, Month 3: number analyzed (Participants) | 214 | 218 | 202 | 226
  hSBA-MenC ≥ 1:8, Month 3 | 213 | 215 | 202 | 226
  hSBA-MenW-135 ≥ 1:4, Month 0: number analyzed (Participants) | 182 | 184 | 190 | 187
  hSBA-MenW-135 ≥ 1:4, Month 0 | 50 | 46 | 54 | 37
  hSBA-MenW-135 ≥ 1:8, Month 0: number analyzed (Participants) | 182 | 184 | 190 | 187
  hSBA-MenW-135 ≥ 1:8, Month 0 | 49 | 44 | 52 | 36
  hSBA-MenW-135 ≥ 1:4, Month 3: number analyzed (Participants) | 201 | 217 | 205 | 204
  hSBA-MenW-135 ≥ 1:4, Month 3 | 197 | 217 | 6 | 3
  hSBA-MenW-135 ≥ 1:8, Month 3: number analyzed (Participants) | 201 | 217 | 205 | 204
  hSBA-MenW-135 ≥ 1:8, Month 3 | 197 | 217 | 4 | 3
  hSBA-MenY ≥ 1:4, Month 0: number analyzed (Participants) | 191 | 192 | 204 | 192
  hSBA-MenY ≥ 1:4, Month 0 | 73 | 73 | 71 | 78
  hSBA-MenY ≥ 1:8, Month 0: number analyzed (Participants) | 191 | 192 | 204 | 192
  hSBA-MenY ≥ 1:8, Month 0 | 73 | 72 | 71 | 77
  hSBA-MenY ≥ 1:4, Month 3: number analyzed (Participants) | 209 | 214 | 204 | 196
  hSBA-MenY ≥ 1:4, Month 3 | 187 | 209 | 11 | 5
  hSBA-MenY ≥ 1:8, Month 3: number analyzed (Participants) | 209 | 214 | 204 | 196
  hSBA-MenY ≥ 1:8, Month 3 | 185 | 209 | 11 | 4

8. Secondary Outcome: hSBA-MenA, hSBA-MenC, hSBA-MenW-135 and hSBA-MenY Antibody Titers
Description: Antibody titers were presented as geometric mean titers (GMTs).
Time Frame: Pre-primary vaccination at Month 0 and one month after final primary vaccination at Month 3
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Nimenrix 3 Group | Nimenrix 2 Group | Menjugate Group | NeisVac-C Group
Number analyzed (Participants) | 214 | 218 | 205 | 226
Titers
  hSBA-MenA, Month 0: number analyzed (Participants) | 164 | 166 | 161 | 166
  hSBA-MenA, Month 0 | 2.8 [2.5 to 3.2] | 2.7 [2.4 to 3] | 3 [2.7 to 3.4] | 2.9 [2.6 to 3.3]
  hSBA-MenA, Month 3: number analyzed (Participants) | 200 | 202 | 172 | 205
  hSBA-MenA, Month 3 | 240.9 [207.8 to 279.3] | 157.2 [131.4 to 188.1] | 2.5 [2.2 to 2.7] | 2.3 [2.2 to 2.5]
  hSBA-MenC, Month 0: number analyzed (Participants) | 181 | 178 | 168 | 185
  hSBA-MenC, Month 0 | 3.9 [3.2 to 4.7] | 3.6 [3 to 4.4] | 4.9 [3.9 to 6.2] | 3.9 [3.2 to 4.7]
  hSBA-MenC, Month 3: number analyzed (Participants) | 214 | 218 | 202 | 226
  hSBA-MenC, Month 3 | 765.6 [647.4 to 905.3] | 1308.3 [1051.7 to 1627.4] | 3188.1 [2645.8 to 3841.5] | 2626.5 [2218.9 to 3109]
  hSBA-MenW-135, Month 0: number analyzed (Participants) | 182 | 184 | 190 | 187
  hSBA-MenW-135, Month 0 | 5 [3.9 to 6.3] | 4.7 [3.8 to 6] | 5 [4 to 6.3] | 3.7 [3.1 to 4.6]
  hSBA-MenW-135, Month 3: number analyzed (Participants) | 201 | 217 | 205 | 204
  hSBA-MenW-135, Month 3 | 190.9 [160 to 227.8] | 753.5 [643.8 to 881.8] | 2.1 [2 to 2.3] | 2.1 [2 to 2.3]
  hSBA-MenY, Month 0: number analyzed (Participants) | 191 | 192 | 204 | 192
  hSBA-MenY, Month 0 | 8 [6.1 to 10.5] | 8 [6.1 to 10.5] | 7.1 [5.5 to 9.2] | 8.1 [6.3 to 10.4]
  hSBA-MenY, Month 3: number analyzed (Participants) | 209 | 214 | 204 | 196
  hSBA-MenY, Month 3 | 66.5 [53.7 to 82.2] | 328.1 [275.8 to 390.2] | 2.4 [2.1 to 2.7] | 2.1 [2 to 2.2]

9. Secondary Outcome: Number of Subjects With hSBA-MenA, hSBA-MenC, hSBA-MenW-135 and hSBA-MenY Antibody Titers Above the Cut-off Values
Description: The cut-off values for hSBA antibody titers were greater than or equal to (≥) 1:4 and ≥ 1:8.
Time Frame: Pre-Booster dose at Month 10 and one month post-Booster dose at Month 11
Population: The analysis was performed on the Booster ATP cohort for immunogenicity, which included all evaluable subjects who used hSBA complement and who complied with the vaccination schedule for Visit 5 (Month 10) and with blood sample schedule for Visit 6 (Month 11).
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix 3 Group | Nimenrix 2 Group | Menjugate Group | NeisVac-C Group
Number analyzed (Participants) | 213 | 221 | 219 | 219
Participants
  hSBA-MenA ≥ 1:4, Month 10: number analyzed (Participants) | 193 | 204 | 188 | 202
  hSBA-MenA ≥ 1:4, Month 10 | 142 | 119 | 28 | 26
  hSBA-MenA ≥ 1:8, Month 10: number analyzed (Participants) | 193 | 204 | 188 | 202
  hSBA-MenA ≥ 1:8, Month 10 | 141 | 119 | 26 | 26
  hSBA-MenA ≥ 1:4, Month 11: number analyzed (Participants) | 212 | 214 | 204 | 205
  hSBA-MenA ≥ 1:4, Month 11 | 210 | 213 | 50 | 55
  hSBA-MenA ≥ 1:8, Month 11: number analyzed (Participants) | 212 | 214 | 204 | 205
  hSBA-MenA ≥ 1:8, Month 11 | 210 | 213 | 50 | 55
  hSBA-MenC ≥ 1:4, Month 10: number analyzed (Participants) | 193 | 208 | 185 | 203
  hSBA-MenC ≥ 1:4, Month 10 | 184 | 198 | 160 | 196
  hSBA-MenC ≥ 1:8, Month 10: number analyzed (Participants) | 193 | 208 | 185 | 203
  hSBA-MenC ≥ 1:8, Month 10 | 184 | 198 | 160 | 196
  hSBA-MenC ≥ 1:4, Month 11: number analyzed (Participants) | 213 | 221 | 216 | 219
  hSBA-MenC ≥ 1:4, Month 11 | 212 | 220 | 216 | 219
  hSBA-MenC ≥ 1:8, Month 11: number analyzed (Participants) | 213 | 221 | 216 | 219
  hSBA-MenC ≥ 1:8, Month 11 | 212 | 220 | 216 | 219
  hSBA-MenW-135 ≥ 1:4, Month 10: number analyzed (Participants) | 198 | 203 | 201 | 210
  hSBA-MenW-135 ≥ 1:4, Month 10 | 196 | 201 | 1 | 6
  hSBA-MenW-135 ≥ 1:8, Month 10: number analyzed (Participants) | 198 | 203 | 201 | 210
  hSBA-MenW-135 ≥ 1:8, Month 10 | 196 | 201 | 1 | 6
  hSBA-MenW-135 ≥ 1:4, Month 11: number analyzed (Participants) | 207 | 218 | 204 | 206
  hSBA-MenW-135 ≥ 1:4, Month 11 | 207 | 218 | 3 | 6
  hSBA-MenW-135 ≥ 1:8, Month 11: number analyzed (Participants) | 207 | 218 | 204 | 206
  hSBA-MenW-135 ≥ 1:8, Month 11 | 207 | 218 | 3 | 6
  hSBA-MenY ≥ 1:4, Month 10: number analyzed (Participants) | 203 | 216 | 219 | 213
  hSBA-MenY ≥ 1:4, Month 10 | 185 | 204 | 6 | 10
  hSBA-MenY ≥ 1:8, Month 10: number analyzed (Participants) | 203 | 216 | 219 | 213
  hSBA-MenY ≥ 1:8, Month 10 | 185 | 204 | 6 | 10
  hSBA-MenY ≥ 1:4, Month 11: number analyzed (Participants) | 206 | 217 | 213 | 217
  hSBA-MenY ≥ 1:4, Month 11 | 206 | 217 | 7 | 12
  hSBA-MenY ≥ 1:8, Month 11: number analyzed (Participants) | 206 | 217 | 213 | 217
  hSBA-MenY ≥ 1:8, Month 11 | 206 | 217 | 7 | 12

10. Secondary Outcome: hSBA-MenA, hSBA-MenC, hSBA-MenW-135 and hSBA-MenY Antibody Titers
Description: Antibody titers were presented as geometric mean titers (GMTs).
Time Frame: Pre-Booster dose at Month 10 and one month post-Booster dose at Month 11
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Nimenrix 3 Group | Nimenrix 2 Group | Menjugate Group | NeisVac-C Group
Number analyzed (Participants) | 213 | 221 | 219 | 219
Titers
  hSBA-MenA, Month 10: number analyzed (Participants) | 193 | 204 | 188 | 202
  hSBA-MenA, Month 10 | 32.0 [24.2 to 42.2] | 14.5 [11.2 to 18.7] | 2.7 [2.4 to 3.0] | 2.7 [2.4 to 3.1]
  hSBA-MenA, Month 11: number analyzed (Participants) | 212 | 214 | 204 | 205
  hSBA-MenA, Month 11 | 1192.7 [978.4 to 1453.9] | 1007.2 [835.7 to 1213.8] | 3.9 [3.3 to 4.6] | 4.2 [3.5 to 5.0]
  hSBA-MenC, Month 10: number analyzed (Participants) | 193 | 208 | 185 | 203
  hSBA-MenC, Month 10 | 116.1 [94.2 to 143.0] | 181.4 [147.3 to 223.4] | 76.8 [58.5 to 100.8] | 213.7 [174.6 to 261.7]
  hSBA-MenC, Month 11: number analyzed (Participants) | 213 | 221 | 216 | 219
  hSBA-MenC, Month 11 | 4411.2 [3654.5 to 5324.6] | 4992.3 [4085.7 to 6100.0] | 5438.2 [4412.4 to 6702.3] | 5542.3 [4765.2 to 6446.2]
  hSBA-MenW-135, Month 10: number analyzed (Participants) | 198 | 203 | 201 | 210
  hSBA-MenW-135, Month 10 | 248.1 [210.4 to 292.6] | 332.4 [287.3 to 384.5] | 2.0 [2.0 to 2.1] | 2.3 [2.0 to 2.6]
  hSBA-MenW-135, Month 11: number analyzed (Participants) | 207 | 218 | 204 | 206
  hSBA-MenW-135, Month 11 | 3944.9 [3419.1 to 4551.7] | 5122.7 [4504.2 to 5826.1] | 2.1 [2.0 to 2.2] | 2.3 [2.1 to 2.7]
  hSBA-MenY, Month 10: number analyzed (Participants) | 203 | 216 | 219 | 213
  hSBA-MenY, Month 10 | 99.8 [80.7 to 123.5] | 140.2 [116.2 to 169.2] | 2.2 [2.0 to 2.4] | 2.4 [2.1 to 2.7]
  hSBA-MenY, Month 11: number analyzed (Participants) | 206 | 217 | 213 | 217
  hSBA-MenY, Month 11 | 2491.5 [2125.8 to 2920.1] | 2954.0 [2497.9 to 3493.3] | 2.3 [2.1 to 2.6] | 2.4 [2.2 to 2.7]

11. Secondary Outcome: Number of Subjects With Anti-pneumococcal Serotypes (Anti-P) Antibody Concentrations Above the Cut-off Values
Description: The cut-off values for anti-1, anti-4, anti-5, anti-6B, anti-7F, anti-9V, anti-14, anti-18C, anti-19F and anti-23F concentrations were greater than or equal to (≥) 0.15 micrograms per milliliter (µg/mL) and ≥ 0.35 µg/mL
Time Frame: Pre-primary vaccination at Month 0 and one month after final primary vaccination at Month 3
Population: The analysis was performed on the Primary ATP cohort for immunogenicity, which included all the evaluable subjects who complied with the vaccination schedule for Visit 1, 2 and 3 (Day 0 to Month 2) and with the blood sample schedule for Visit 4 (Month 3), as assessed for a randomized subset of 25% of subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix 3 Group | Nimenrix 2 Group | Menjugate Group | NeisVac-C Group
Number analyzed (Participants) | 98 | 104 | 95 | 103
Participants
  Anti-1 ≥ 0.15 µg/mL, Month 0: number analyzed (Participants) | 98 | 92 | 90 | 97
  Anti-1 ≥ 0.15 µg/mL, Month 0 | 18 | 15 | 17 | 18
  Anti-1 ≥ 0.35 µg/mL, Month 0: number analyzed (Participants) | 98 | 92 | 90 | 97
  Anti-1 ≥ 0.35 µg/mL, Month 0 | 3 | 9 | 8 | 8
  Anti-1 ≥ 0.15 µg/mL, Month 3: number analyzed (Participants) | 96 | 104 | 93 | 103
  Anti-1 ≥ 0.15 µg/mL, Month 3 | 96 | 102 | 93 | 103
  Anti-1 ≥ 0.35 µg/mL, Month 3: number analyzed (Participants) | 96 | 104 | 93 | 103
  Anti-1 ≥ 0.35 µg/mL, Month 3 | 93 | 95 | 89 | 91
  Anti-4 ≥ 0.15 µg/mL, Month 0: number analyzed (Participants) | 98 | 93 | 92 | 95
  Anti-4 ≥ 0.15 µg/mL, Month 0 | 11 | 11 | 13 | 12
  Anti-4 ≥ 0.35 µg/mL, Month 0: number analyzed (Participants) | 98 | 93 | 92 | 95
  Anti-4 ≥ 0.35 µg/mL, Month 0 | 2 | 2 | 2 | 1
  Anti-4 ≥ 0.15 µg/mL, Month 3: number analyzed (Participants) | 96 | 104 | 95 | 103
  Anti-4 ≥ 0.15 µg/mL, Month 3 | 96 | 102 | 95 | 103
  Anti-4 ≥ 0.35 µg/mL, Month 3: number analyzed (Participants) | 96 | 104 | 95 | 103
  Anti-4 ≥ 0.35 µg/mL, Month 3 | 94 | 99 | 93 | 99
  Anti-5 ≥ 0.15 µg/mL, Month 0: number analyzed (Participants) | 97 | 92 | 91 | 96
  Anti-5 ≥ 0.15 µg/mL, Month 0 | 42 | 32 | 39 | 33
  Anti-5 ≥ 0.35 µg/mL, Month 0: number analyzed (Participants) | 97 | 92 | 91 | 96
  Anti-5 ≥ 0.35 µg/mL, Month 0 | 10 | 5 | 9 | 14
  Anti-5 ≥ 0.15 µg/mL, Month 3: number analyzed (Participants) | 96 | 104 | 93 | 103
  Anti-5 ≥ 0.15 µg/mL, Month 3 | 95 | 102 | 93 | 101
  Anti-5 ≥ 0.35 µg/mL, Month 3: number analyzed (Participants) | 96 | 104 | 93 | 103
  Anti-5 ≥ 0.35 µg/mL, Month 3 | 84 | 86 | 80 | 92
  Anti-6B ≥ 0.15 µg/mL, Month 0: number analyzed (Participants) | 97 | 92 | 91 | 96
  Anti-6B ≥ 0.15 µg/mL, Month 0 | 55 | 42 | 41 | 50
  Anti-6B ≥ 0.35 µg/mL, Month 0: number analyzed (Participants) | 97 | 92 | 91 | 96
  Anti-6B ≥ 0.35 µg/mL, Month 0 | 27 | 19 | 20 | 26
  Anti-6B ≥ 0.15 µg/mL, Month 3: number analyzed (Participants) | 96 | 104 | 93 | 103
  Anti-6B ≥ 0.15 µg/mL, Month 3 | 88 | 95 | 88 | 90
  Anti-6B ≥ 0.35 µg/mL, Month 3: number analyzed (Participants) | 96 | 104 | 93 | 103
  Anti-6B ≥ 0.35 µg/mL, Month 3 | 71 | 82 | 75 | 81
  Anti-7F ≥ 0.15 µg/mL, Month 0: number analyzed (Participants) | 98 | 92 | 92 | 96
  Anti-7F ≥ 0.15 µg/mL, Month 0 | 38 | 43 | 44 | 49
  Anti-7F ≥ 0.35 µg/mL, Month 0: number analyzed (Participants) | 98 | 92 | 92 | 96
  Anti-7F ≥ 0.35 µg/mL, Month 0 | 13 | 18 | 20 | 16
  Anti-7F ≥ 0.15 µg/mL, Month 3: number analyzed (Participants) | 96 | 104 | 93 | 103
  Anti-7F ≥ 0.15 µg/mL, Month 3 | 96 | 102 | 93 | 103
  Anti-7F ≥ 0.35 µg/mL, Month 3: number analyzed (Participants) | 96 | 104 | 93 | 103
  Anti-7F ≥ 0.35 µg/mL, Month 3 | 94 | 99 | 93 | 103
  Anti-9V ≥ 0.15 µg/mL, Month 0: number analyzed (Participants) | 97 | 93 | 92 | 96
  Anti-9V ≥ 0.15 µg/mL, Month 0 | 38 | 44 | 35 | 43
  Anti-9V ≥ 0.35 µg/mL, Month 0: number analyzed (Participants) | 97 | 93 | 92 | 96
  Anti-9V ≥ 0.35 µg/mL, Month 0 | 9 | 18 | 12 | 16
  Anti-9V ≥ 0.15 µg/mL, Month 3: number analyzed (Participants) | 96 | 104 | 93 | 103
  Anti-9V ≥ 0.15 µg/mL, Month 3 | 94 | 102 | 90 | 103
  Anti-9V ≥ 0.35 µg/mL, Month 3: number analyzed (Participants) | 96 | 104 | 93 | 103
  Anti-9V ≥ 0.35 µg/mL, Month 3 | 92 | 99 | 88 | 99
  Anti-14 ≥ 0.15 µg/mL, Month 0: number analyzed (Participants) | 97 | 92 | 90 | 95
  Anti-14 ≥ 0.15 µg/mL, Month 0 | 72 | 69 | 74 | 80
  Anti-14 ≥ 0.35 µg/mL, Month 0: number analyzed (Participants) | 97 | 92 | 90 | 95
  Anti-14 ≥ 0.35 µg/mL, Month 0 | 53 | 57 | 57 | 67
  Anti-14 ≥ 0.15 µg/mL, Month 3: number analyzed (Participants) | 96 | 103 | 95 | 103
  Anti-14 ≥ 0.15 µg/mL, Month 3 | 96 | 103 | 95 | 103
  Anti-14 ≥ 0.35 µg/mL, Month 3: number analyzed (Participants) | 96 | 103 | 95 | 103
  Anti-14 ≥ 0.35 µg/mL, Month 3 | 96 | 103 | 95 | 103
  Anti-18C ≥ 0.15 µg/mL, Month 0: number analyzed (Participants) | 96 | 93 | 91 | 94
  Anti-18C ≥ 0.15 µg/mL, Month 0 | 30 | 44 | 45 | 43
  Anti-18C ≥ 0.35 µg/mL, Month 0: number analyzed (Participants) | 96 | 93 | 91 | 94
  Anti-18C ≥ 0.35 µg/mL, Month 0 | 14 | 18 | 20 | 10
  Anti-18C ≥ 0.15 µg/mL, Month 3: number analyzed (Participants) | 96 | 103 | 94 | 103
  Anti-18C ≥ 0.15 µg/mL, Month 3 | 96 | 101 | 93 | 103
  Anti-18C ≥ 0.35 µg/mL, Month 3: number analyzed (Participants) | 96 | 103 | 94 | 103
  Anti-18C ≥ 0.35 µg/mL, Month 3 | 90 | 100 | 89 | 101
  Anti-19F ≥ 0.15 µg/mL, Month 0: number analyzed (Participants) | 96 | 93 | 91 | 96
  Anti-19F ≥ 0.15 µg/mL, Month 0 | 41 | 61 | 51 | 53
  Anti-19F ≥ 0.35 µg/mL, Month 0: number analyzed (Participants) | 96 | 93 | 91 | 96
  Anti-19F ≥ 0.35 µg/mL, Month 0 | 21 | 30 | 27 | 23
  Anti-19F ≥ 0.15 µg/mL, Month 3: number analyzed (Participants) | 96 | 104 | 95 | 103
  Anti-19F ≥ 0.15 µg/mL, Month 3 | 94 | 100 | 94 | 102
  Anti-19F ≥ 0.35 µg/mL, Month 3: number analyzed (Participants) | 96 | 104 | 95 | 103
  Anti-19F ≥ 0.35 µg/mL, Month 3 | 92 | 94 | 90 | 99
  Anti-23F ≥ 0.15 µg/mL, Month 0: number analyzed (Participants) | 97 | 92 | 90 | 96
  Anti-23F ≥ 0.15 µg/mL, Month 0 | 37 | 38 | 29 | 40
  Anti-23F ≥ 0.35 µg/mL, Month 0: number analyzed (Participants) | 97 | 92 | 90 | 96
  Anti-23F ≥ 0.35 µg/mL, Month 0 | 16 | 13 | 13 | 18
  Anti-23F ≥ 0.15 µg/mL, Month 3: number analyzed (Participants) | 95 | 104 | 94 | 103
  Anti-23F ≥ 0.15 µg/mL, Month 3 | 90 | 99 | 91 | 98
  Anti-23F ≥ 0.35 µg/mL, Month 3: number analyzed (Participants) | 95 | 104 | 94 | 103
  Anti-23F ≥ 0.35 µg/mL, Month 3 | 83 | 83 | 77 | 86

12. Secondary Outcome: Anti-pneumococcal Serotypes Antibody Concentrations
Description: Anti-1, anti-4, anti-5, anti-6B, anti-7F, anti-9V, anti-14, anti-18C, anti-19F and anti-23F antibody concentrations were presented as geometric mean concentrations (GMCs) and expressed in µg/mL.
Time Frame: Pre-primary vaccination at Month 0 and one month after final primary vaccination at Month 3
Population: as for outcome 11
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | Nimenrix 3 Group | Nimenrix 2 Group | Menjugate Group | NeisVac-C Group
Number analyzed (Participants) | 98 | 104 | 95 | 103
µg/mL
  Anti-1, Month 0: number analyzed (Participants) | 98 | 92 | 90 | 97
  Anti-1, Month 0 | 0.09 [0.08 to 0.10] | 0.10 [0.09 to 0.12] | 0.10 [0.09 to 0.12] | 0.10 [0.09 to 0.11]
  Anti-1, Month 3: number analyzed (Participants) | 96 | 104 | 93 | 103
  Anti-1, Month 3 | 1.36 [1.15 to 1.62] | 1.13 [0.96 to 1.34] | 1.26 [1.06 to 1.50] | 1.02 [0.88 to 1.18]
  Anti-4, Month 0: number analyzed (Participants) | 98 | 93 | 92 | 95
  Anti-4, Month 0 | 0.09 [0.08 to 0.09] | 0.09 [0.08 to 0.09] | 0.09 [0.08 to 0.10] | 0.09 [0.08 to 0.09]
  Anti-4, Month 3: number analyzed (Participants) | 96 | 104 | 95 | 103
  Anti-4, Month 3 | 1.84 [1.58 to 2.15] | 1.56 [1.31 to 1.86] | 1.77 [1.50 to 2.10] | 1.60 [1.37 to 1.85]
  Anti-5, Month 0: number analyzed (Participants) | 97 | 92 | 91 | 96
  Anti-5, Month 0 | 0.13 [0.11 to 0.15] | 0.12 [0.10 to 0.13] | 0.13 [0.11 to 0.15] | 0.12 [0.11 to 0.15]
  Anti-5, Month 3: number analyzed (Participants) | 96 | 104 | 93 | 103
  Anti-5, Month 3 | 0.82 [0.71 to 0.95] | 0.70 [0.61 to 0.81] | 0.77 [0.66 to 0.89] | 0.74 [0.65 to 0.85]
  Anti-6B, Month 0: number analyzed (Participants) | 97 | 92 | 91 | 96
  Anti-6B, Month 0 | 0.18 [0.15 to 0.21] | 0.15 [0.13 to 0.19] | 0.15 [0.13 to 0.19] | 0.18 [0.15 to 0.22]
  Anti-6B, Month 3: number analyzed (Participants) | 96 | 104 | 93 | 103
  Anti-6B, Month 3 | 0.79 [0.62 to 1.00] | 0.90 [0.71 to 1.14] | 1.08 [0.84 to 1.38] | 0.86 [0.67 to 1.12]
  Anti-7F, Month 0: number analyzed (Participants) | 98 | 92 | 92 | 96
  Anti-7F, Month 0 | 0.13 [0.11 to 0.16] | 0.17 [0.13 to 0.21] | 0.16 [0.13 to 0.20] | 0.15 [0.13 to 0.18]
  Anti-7F, Month 3: number analyzed (Participants) | 96 | 104 | 93 | 103
  Anti-7F, Month 3 | 1.91 [1.63 to 2.23] | 1.84 [1.56 to 2.18] | 2.13 [1.82 to 2.49] | 1.87 [1.62 to 2.15]
  Anti-9V, Month 0: number analyzed (Participants) | 97 | 93 | 92 | 96
  Anti-9V, Month 0 | 0.13 [0.11 to 0.15] | 0.15 [0.13 to 0.18] | 0.13 [0.11 to 0.15] | 0.14 [0.12 to 0.17]
  Anti-9V, Month 3: number analyzed (Participants) | 96 | 104 | 93 | 103
  Anti-9V, Month 3 | 1.31 [1.10 to 1.56] | 1.12 [0.97 to 1.29] | 1.22 [1.02 to 1.46] | 1.21 [1.07 to 1.38]
  Anti-14, Month 0: number analyzed (Participants) | 97 | 92 | 90 | 95
  Anti-14, Month 0 | 0.50 [0.37 to 0.67] | 0.61 [0.44 to 0.85] | 0.59 [0.44 to 0.79] | 0.74 [0.56 to 0.99]
  Anti-14, Month 3: number analyzed (Participants) | 96 | 103 | 95 | 103
  Anti-14, Month 3 | 7.55 [6.40 to 8.90] | 7.40 [6.35 to 8.62] | 8.51 [7.09 to 10.22] | 6.04 [5.04 to 7.24]
  Anti-18C, Month 0: number analyzed (Participants) | 96 | 93 | 91 | 94
  Anti-18C, Month 0 | 0.13 [0.11 to 0.16] | 0.16 [0.13 to 0.20] | 0.17 [0.14 to 0.21] | 0.14 [0.12 to 0.16]
  Anti-18C, Month 3: number analyzed (Participants) | 96 | 103 | 94 | 103
  Anti-18C, Month 3 | 2.14 [1.74 to 2.64] | 1.77 [1.47 to 2.13] | 2.39 [1.96 to 2.93] | 2.80 [2.40 to 3.27]
  Anti-19F, Month 0: number analyzed (Participants) | 96 | 93 | 91 | 96
  Anti-19F, Month 0 | 0.15 [0.13 to 0.19] | 0.23 [0.19 to 0.28] | 0.20 [0.16 to 0.25] | 0.19 [0.15 to 0.23]
  Anti-19F, Month 3: number analyzed (Participants) | 96 | 104 | 95 | 103
  Anti-19F, Month 3 | 3.01 [2.37 to 3.82] | 2.60 [2.01 to 3.35] | 2.89 [2.26 to 3.69] | 2.85 [2.29 to 3.54]
  Anti-23F, Month 0: number analyzed (Participants) | 97 | 92 | 90 | 96
  Anti-23F, Month 0 | 0.14 [0.11 to 0.16] | 0.14 [0.11 to 0.17] | 0.13 [0.11 to 0.15] | 0.15 [0.12 to 0.17]
  Anti-23F, Month 3: number analyzed (Participants) | 95 | 104 | 94 | 103
  Anti-23F, Month 3 | 0.96 [0.78 to 1.18] | 0.85 [0.69 to 1.06] | 1.08 [0.86 to 1.36] | 0.94 [0.77 to 1.16]

13. Secondary Outcome: Number of Subjects With Anti-pneumococcal Serotypes Antibody Concentrations Above the Cut-off Values
Description: The cut-off values for anti-1, anti-4, anti-5, anti-6B, anti-7F, anti-9V, anti-14, anti-18C, anti-19F and anti-23F concentrations were ≥ 0.15 µg/mL and ≥ 0.35 µg/mL
Time Frame: Pre-Booster dose at Month 10 and one month post-Booster dose at Month 11
Population: The analysis was performed on the Booster ATP cohort for immunogenicity, which included all the evaluable subjects who complied with the vaccination schedule for Visit 5 (Month 10) and with blood sample schedule for Visit 6 (Month 11), as assessed for a randomized subset of 25% of subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix 3 Group | Nimenrix 2 Group | Menjugate Group | NeisVac-C Group
Number analyzed (Participants) | 104 | 107 | 106 | 110
Participants
  Anti-1 ≥ 0.15 µg/mL, Month 10: number analyzed (Participants) | 102 | 107 | 106 | 109
  Anti-1 ≥ 0.15 µg/mL, Month 10 | 65 | 64 | 72 | 57
  Anti-1 ≥ 0.35 µg/mL, Month 10: number analyzed (Participants) | 102 | 107 | 106 | 109
  Anti-1 ≥ 0.35 µg/mL, Month 10 | 21 | 20 | 24 | 10
  Anti-1 ≥ 0.15 µg/mL, Month 11: number analyzed (Participants) | 104 | 107 | 100 | 103
  Anti-1 ≥ 0.15 µg/mL, Month 11 | 104 | 106 | 99 | 103
  Anti-1 ≥ 0.35 µg/mL, Month 11: number analyzed (Participants) | 104 | 107 | 100 | 103
  Anti-1 ≥ 0.35 µg/mL, Month 11 | 102 | 104 | 97 | 101
  Anti-4 ≥ 0.15 µg/mL, Month 10: number analyzed (Participants) | 102 | 107 | 106 | 110
  Anti-4 ≥ 0.15 µg/mL, Month 10 | 83 | 87 | 91 | 94
  Anti-4 ≥ 0.35 µg/mL, Month 10: number analyzed (Participants) | 102 | 107 | 106 | 110
  Anti-4 ≥ 0.35 µg/mL, Month 10 | 38 | 35 | 48 | 30
  Anti-4 ≥ 0.15 µg/mL, Month 11: number analyzed (Participants) | 104 | 107 | 100 | 104
  Anti-4 ≥ 0.15 µg/mL, Month 11 | 104 | 107 | 100 | 104
  Anti-4 ≥ 0.35 µg/mL, Month 11: number analyzed (Participants) | 104 | 107 | 100 | 104
  Anti-4 ≥ 0.35 µg/mL, Month 11 | 104 | 107 | 99 | 104
  Anti-5 ≥ 0.15 µg/mL, Month 10: number analyzed (Participants) | 102 | 107 | 106 | 110
  Anti-5 ≥ 0.15 µg/mL, Month 10 | 90 | 91 | 94 | 93
  Anti-5 ≥ 0.35 µg/mL, Month 10: number analyzed (Participants) | 102 | 107 | 106 | 110
  Anti-5 ≥ 0.35 µg/mL, Month 10 | 44 | 43 | 48 | 43
  Anti-5 ≥ 0.15 µg/mL, Month 11: number analyzed (Participants) | 101 | 104 | 98 | 101
  Anti-5 ≥ 0.15 µg/mL, Month 11 | 101 | 104 | 98 | 101
  Anti-5 ≥ 0.35 µg/mL, Month 11: number analyzed (Participants) | 101 | 104 | 98 | 101
  Anti-5 ≥ 0.35 µg/mL, Month 11 | 92 | 96 | 95 | 96
  Anti-6B ≥ 0.15 µg/mL, Month 10: number analyzed (Participants) | 99 | 106 | 106 | 108
  Anti-6B ≥ 0.15 µg/mL, Month 10 | 96 | 104 | 104 | 103
  Anti-6B ≥ 0.35 µg/mL, Month 10: number analyzed (Participants) | 99 | 106 | 106 | 108
  Anti-6B ≥ 0.35 µg/mL, Month 10 | 71 | 84 | 83 | 83
  Anti-6B ≥ 0.15 µg/mL, Month 11: number analyzed (Participants) | 104 | 107 | 100 | 104
  Anti-6B ≥ 0.15 µg/mL, Month 11 | 103 | 106 | 100 | 104
  Anti-6B ≥ 0.35 µg/mL, Month 11: number analyzed (Participants) | 104 | 107 | 100 | 104
  Anti-6B ≥ 0.35 µg/mL, Month 11 | 103 | 105 | 100 | 104
  Anti-7F ≥ 0.15 µg/mL, Month 10: number analyzed (Participants) | 102 | 107 | 106 | 110
  Anti-7F ≥ 0.15 µg/mL, Month 10 | 98 | 103 | 106 | 104
  Anti-7F ≥ 0.35 µg/mL, Month 10: number analyzed (Participants) | 102 | 107 | 106 | 110
  Anti-7F ≥ 0.35 µg/mL, Month 10 | 76 | 78 | 75 | 78
  Anti-7F ≥ 0.15 µg/mL, Month 11: number analyzed (Participants) | 104 | 107 | 100 | 104
  Anti-7F ≥ 0.15 µg/mL, Month 11 | 104 | 107 | 100 | 104
  Anti-7F ≥ 0.35 µg/mL, Month 11: number analyzed (Participants) | 104 | 107 | 100 | 104
  Anti-7F ≥ 0.35 µg/mL, Month 11 | 104 | 107 | 100 | 104
  Anti-9V ≥ 0.15 µg/mL, Month 10: number analyzed (Participants) | 102 | 107 | 105 | 109
  Anti-9V ≥ 0.15 µg/mL, Month 10 | 81 | 82 | 88 | 89
  Anti-9V ≥ 0.35 µg/mL, Month 10: number analyzed (Participants) | 102 | 107 | 105 | 109
  Anti-9V ≥ 0.35 µg/mL, Month 10 | 42 | 30 | 43 | 33
  Anti-9V ≥ 0.15 µg/mL, Month 11: number analyzed (Participants) | 104 | 107 | 100 | 104
  Anti-9V ≥ 0.15 µg/mL, Month 11 | 104 | 107 | 100 | 104
  Anti-9V ≥ 0.35 µg/mL, Month 11: number analyzed (Participants) | 104 | 107 | 100 | 104
  Anti-9V ≥ 0.35 µg/mL, Month 11 | 102 | 105 | 99 | 102
  Anti-14 ≥ 0.15 µg/mL, Month 10: number analyzed (Participants) | 102 | 107 | 106 | 109
  Anti-14 ≥ 0.15 µg/mL, Month 10 | 102 | 106 | 106 | 106
  Anti-14 ≥ 0.35 µg/mL, Month 10: number analyzed (Participants) | 102 | 107 | 106 | 109
  Anti-14 ≥ 0.35 µg/mL, Month 10 | 100 | 103 | 99 | 103
  Anti-14 ≥ 0.15 µg/mL, Month 11: number analyzed (Participants) | 104 | 107 | 100 | 104
  Anti-14 ≥ 0.15 µg/mL, Month 11 | 104 | 107 | 100 | 104
  Anti-14 ≥ 0.35 µg/mL, Month 11: number analyzed (Participants) | 104 | 107 | 100 | 104
  Anti-14 ≥ 0.35 µg/mL, Month 11 | 104 | 107 | 100 | 104
  Anti-18C ≥ 0.15 µg/mL, Month 10: number analyzed (Participants) | 101 | 107 | 106 | 110
  Anti-18C ≥ 0.15 µg/mL, Month 10 | 82 | 89 | 97 | 101
  Anti-18C ≥ 0.35 µg/mL, Month 10: number analyzed (Participants) | 101 | 107 | 106 | 110
  Anti-18C ≥ 0.35 µg/mL, Month 10 | 45 | 50 | 54 | 58
  Anti-18C ≥ 0.15 µg/mL, Month 11: number analyzed (Participants) | 103 | 107 | 100 | 104
  Anti-18C ≥ 0.15 µg/mL, Month 11 | 103 | 107 | 100 | 104
  Anti-18C ≥ 0.35 µg/mL, Month 11: number analyzed (Participants) | 103 | 107 | 100 | 104
  Anti-18C ≥ 0.35 µg/mL, Month 11 | 103 | 106 | 100 | 104
  Anti-19F ≥ 0.15 µg/mL, Month 10: number analyzed (Participants) | 102 | 107 | 106 | 109
  Anti-19F ≥ 0.15 µg/mL, Month 10 | 102 | 107 | 106 | 107
  Anti-19F ≥ 0.35 µg/mL, Month 10: number analyzed (Participants) | 102 | 107 | 106 | 109
  Anti-19F ≥ 0.35 µg/mL, Month 10 | 96 | 98 | 103 | 102
  Anti-19F ≥ 0.15 µg/mL, Month 11: number analyzed (Participants) | 104 | 107 | 100 | 104
  Anti-19F ≥ 0.15 µg/mL, Month 11 | 104 | 107 | 100 | 104
  Anti-19F ≥ 0.35 µg/mL, Month 11: number analyzed (Participants) | 104 | 107 | 100 | 104
  Anti-19F ≥ 0.35 µg/mL, Month 11 | 104 | 107 | 100 | 104
  Anti-23F ≥ 0.15 µg/mL, Month 10: number analyzed (Participants) | 102 | 107 | 106 | 110
  Anti-23F ≥ 0.15 µg/mL, Month 10 | 94 | 103 | 102 | 101
  Anti-23F ≥ 0.35 µg/mL, Month 10: number analyzed (Participants) | 102 | 107 | 106 | 110
  Anti-23F ≥ 0.35 µg/mL, Month 10 | 58 | 61 | 63 | 63
  Anti-23F ≥ 0.15 µg/mL, Month 11: number analyzed (Participants) | 101 | 106 | 98 | 104
  Anti-23F ≥ 0.15 µg/mL, Month 11 | 101 | 106 | 98 | 104
  Anti-23F ≥ 0.35 µg/mL, Month 11: number analyzed (Participants) | 101 | 106 | 98 | 104
  Anti-23F ≥ 0.35 µg/mL, Month 11 | 101 | 106 | 98 | 104

14. Secondary Outcome: Anti-pneumococcal Serotypes Antibody Concentrations
Description: as for outcome 12
Time Frame: Pre-Booster dose at Month 10 and one month post-Booster dose at Month 11
Population: as for outcome 13
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | Nimenrix 3 Group | Nimenrix 2 Group | Menjugate Group | NeisVac-C Group
Number analyzed (Participants) | 104 | 107 | 106 | 110
µg/mL
  Anti-1, Month 10: number analyzed (Participants) | 102 | 107 | 106 | 109
  Anti-1, Month 10 | 0.19 [0.16 to 0.22] | 0.17 [0.15 to 0.20] | 0.20 [0.17 to 0.23] | 0.15 [0.13 to 0.17]
  Anti-1, Month 11: number analyzed (Participants) | 104 | 107 | 100 | 103
  Anti-1, Month 11 | 2.03 [1.72 to 2.41] | 1.67 [1.39 to 2.01] | 2.18 [1.81 to 2.64] | 1.72 [1.46 to 2.03]
  Anti-4, Month 10: number analyzed (Participants) | 102 | 107 | 106 | 110
  Anti-4, Month 10 | 0.27 [0.23 to 0.32] | 0.27 [0.23 to 0.32] | 0.31 [0.27 to 0.37] | 0.25 [0.22 to 0.28]
  Anti-4, Month 11: number analyzed (Participants) | 104 | 107 | 100 | 104
  Anti-4, Month 11 | 2.42 [2.11 to 2.78] | 2.16 [1.86 to 2.51] | 2.86 [2.46 to 3.34] | 2.12 [1.87 to 2.40]
  Anti-5, Month 10: number analyzed (Participants) | 102 | 107 | 106 | 110
  Anti-5, Month 10 | 0.32 [0.27 to 0.37] | 0.28 [0.24 to 0.32] | 0.30 [0.26 to 0.35] | 0.27 [0.23 to 0.30]
  Anti-5, Month 11: number analyzed (Participants) | 101 | 104 | 98 | 101
  Anti-5, Month 11 | 0.89 [0.78 to 1.02] | 0.87 [0.76 to 1.00] | 0.95 [0.83 to 1.09] | 0.84 [0.74 to 0.97]
  Anti-6B, Month 10: number analyzed (Participants) | 99 | 106 | 106 | 108
  Anti-6B, Month 10 | 0.62 [0.52 to 0.73] | 0.64 [0.54 to 0.76] | 0.68 [0.58 to 0.80] | 0.59 [0.51 to 0.69]
  Anti-6B, Month 11: number analyzed (Participants) | 104 | 107 | 100 | 104
  Anti-6B, Month 11 | 2.91 [2.49 to 3.41] | 3.02 [2.57 to 3.56] | 3.70 [3.18 to 4.29] | 3.20 [2.79 to 3.68]
  Anti-7F, Month 10: number analyzed (Participants) | 102 | 107 | 106 | 110
  Anti-7F, Month 10 | 0.50 [0.44 to 0.57] | 0.52 [0.45 to 0.61] | 0.57 [0.50 to 0.66] | 0.46 [0.40 to 0.52]
  Anti-7F, Month 11: number analyzed (Participants) | 104 | 107 | 100 | 104
  Anti-7F, Month 11 | 2.89 [2.53 to 3.30] | 2.88 [2.51 to 3.31] | 3.38 [2.94 to 3.89] | 2.78 [2.43 to 3.17]
  Anti-9V, Month 10: number analyzed (Participants) | 102 | 107 | 105 | 109
  Anti-9V, Month 10 | 0.27 [0.23 to 0.33] | 0.23 [0.20 to 0.27] | 0.28 [0.24 to 0.32] | 0.25 [0.22 to 0.28]
  Anti-9V, Month 11: number analyzed (Participants) | 104 | 107 | 100 | 104
  Anti-9V, Month 11 | 1.49 [1.30 to 1.70] | 1.31 [1.15 to 1.49] | 1.47 [1.27 to 1.71] | 1.33 [1.18 to 1.49]
  Anti-14, Month 10: number analyzed (Participants) | 102 | 107 | 106 | 109
  Anti-14, Month 10 | 1.69 [1.39 to 2.05] | 1.64 [1.37 to 1.97] | 1.74 [1.46 to 2.09] | 1.42 [1.18 to 1.70]
  Anti-14, Month 11: number analyzed (Participants) | 104 | 107 | 100 | 104
  Anti-14, Month 11 | 8.51 [7.20 to 10.07] | 7.63 [6.62 to 8.79] | 9.75 [8.36 to 11.38] | 7.94 [6.85 to 9.20]
  Anti-18C, Month 10: number analyzed (Participants) | 101 | 107 | 106 | 110
  Anti-18C, Month 10 | 0.33 [0.27 to 0.40] | 0.33 [0.28 to 0.39] | 0.39 [0.33 to 0.46] | 0.38 [0.33 to 0.44]
  Anti-18C, Month 11: number analyzed (Participants) | 103 | 107 | 100 | 104
  Anti-18C, Month 11 | 2.30 [2.00 to 2.64] | 2.10 [1.84 to 2.39] | 3.08 [2.65 to 3.58] | 2.78 [2.44 to 3.17]
  Anti-19F, Month 10: number analyzed (Participants) | 102 | 107 | 106 | 109
  Anti-19F, Month 10 | 1.22 [1.04 to 1.45] | 1.26 [1.05 to 1.52] | 1.34 [1.13 to 1.59] | 1.10 [0.94 to 1.29]
  Anti-19F, Month 11: number analyzed (Participants) | 104 | 107 | 100 | 104
  Anti-19F, Month 11 | 9.55 [8.23 to 11.09] | 8.06 [6.88 to 9.46] | 9.74 [8.20 to 11.58] | 8.43 [7.35 to 9.66]
  Anti-23F, Month 10: number analyzed (Participants) | 102 | 107 | 106 | 110
  Anti-23F, Month 10 | 0.39 [0.34 to 0.46] | 0.45 [0.39 to 0.53] | 0.47 [0.40 to 0.56] | 0.41 [0.35 to 0.48]
  Anti-23F, Month 11: number analyzed (Participants) | 101 | 106 | 98 | 104
  Anti-23F, Month 11 | 3.74 [3.23 to 4.34] | 3.73 [3.19 to 4.35] | 4.24 [3.60 to 5.00] | 3.73 [3.30 to 4.21]

15. Secondary Outcome: Number of Subjects With Anti-diphtheria (Anti-D) and Anti-tetanus (Anti-T) Concentrations ≥ the Cut-off Value
Description: The cut-off value for anti-D and anti-T concentrations was greater than or equal to (≥) 0.1 IU/mL
Time Frame: Pre-primary vaccination at Month 0 and one month after final primary vaccination at Month 3
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix 3 Group | Nimenrix 2 Group | Menjugate Group | NeisVac-C Group
Number analyzed (Participants) | 117 | 113 | 123 | 115
Participants
  Anti-D, Month 0: number analyzed (Participants) | 116 | 106 | 117 | 110
  Anti-D, Month 0 | 37 | 43 | 56 | 39
  Anti-D, Month 3 | 117 | 113 | 123 | 115
  Anti-T, Month 0: number analyzed (Participants) | 116 | 107 | 116 | 111
  Anti-T, Month 0 | 104 | 91 | 107 | 91
  Anti-T, Month 3: number analyzed (Participants) | 117 | 113 | 123 | 114
  Anti-T, Month 3 | 117 | 113 | 123 | 114

16. Secondary Outcome: Anti-D and Anti-T Antibody Concentrations
Description: Antibody concentrations were presented as geometric mean concentrations (GMCs) and expressed in international units per milliliter (IU/mL).
Time Frame: Pre-primary vaccination at Month 0 and one month after final primary vaccination at Month 3
Population: as for outcome 11
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Nimenrix 3 Group | Nimenrix 2 Group | Menjugate Group | NeisVac-C Group
Number analyzed (Participants) | 117 | 113 | 123 | 115
IU/mL
  Anti-D, Month 0: number analyzed (Participants) | 116 | 106 | 117 | 110
  Anti-D, Month 0 | 0.092 [0.077 to 0.11] | 0.098 [0.082 to 0.117] | 0.133 [0.108 to 0.165] | 0.093 [0.078 to 0.112]
  Anti-D, Month 3 | 2.171 [1.893 to 2.49] | 2.64 [2.274 to 3.065] | 3.005 [2.657 to 3.4] | 2.488 [2.169 to 2.855]
  Anti-T, Month 0: number analyzed (Participants) | 116 | 107 | 116 | 111
  Anti-T, Month 0 | 0.484 [0.393 to 0.596] | 0.496 [0.388 to 0.636] | 0.727 [0.581 to 0.909] | 0.5 [0.387 to 0.647]
  Anti-T, Month 3: number analyzed (Participants) | 117 | 113 | 123 | 114
  Anti-T, Month 3 | 3.137 [2.79 to 3.527] | 3.37 [2.98 to 3.811] | 2.847 [2.523 to 3.212] | 4.339 [3.833 to 4.912]

17. Secondary Outcome: Number of Subjects With Anti-D and Anti-T Antibody Concentrations ≥ the Cut-off Value
Description: The cut-off value for anti-D and anti-T concentrations was greater than or equal to (≥) 0.1 IU/mL
Time Frame: Pre-Booster dose at Month 10 and one month post-Booster dose at Month 11
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix 3 Group | Nimenrix 2 Group | Menjugate Group | NeisVac-C Group
Number analyzed (Participants) | 116 | 112 | 119 | 118
Participants
  Anti-D, Month 10: number analyzed (Participants) | 114 | 112 | 119 | 117
  Anti-D, Month 10 | 98 | 98 | 116 | 113
  Anti-D, Month 11: number analyzed (Participants) | 116 | 111 | 118 | 118
  Anti-D, Month 11 | 116 | 111 | 118 | 118
  Anti-T, Month 10: number analyzed (Participants) | 114 | 112 | 119 | 117
  Anti-T, Month 10 | 114 | 111 | 118 | 117
  Anti-T, Month 11: number analyzed (Participants) | 116 | 111 | 118 | 118
  Anti-T, Month 11 | 116 | 111 | 118 | 118

18. Secondary Outcome: Anti-D and Anti-T Antibody Concentrations
Description: as for outcome 16
Time Frame: Pre-Booster dose at Month 10 and one month post-Booster dose at Month 11
Population: as for outcome 13
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Nimenrix 3 Group | Nimenrix 2 Group | Menjugate Group | NeisVac-C Group
Number analyzed (Participants) | 116 | 112 | 119 | 118
IU/mL
  Anti-D, Month 10: number analyzed (Participants) | 114 | 112 | 119 | 117
  Anti-D, Month 10 | 0.292 [0.246 to 0.348] | 0.325 [0.272 to 0.389] | 0.507 [0.433 to 0.594] | 0.379 [0.327 to 0.440]
  Anti-D, Month 11: number analyzed (Participants) | 116 | 111 | 118 | 118
  Anti-D, Month 11 | 5.032 [4.337 to 5.838] | 5.438 [4.600 to 6.430] | 9.078 [7.959 to 10.354] | 6.437 [5.589 to 7.413]
  Anti-T, Month 10: number analyzed (Participants) | 114 | 112 | 119 | 117
  Anti-T, Month 10 | 0.832 [0.739 to 0.937] | 0.780 [0.677 to 0.898] | 0.684 [0.590 to 0.793] | 0.956 [0.835 to 1.094]
  Anti-T, Month 11: number analyzed (Participants) | 116 | 111 | 118 | 118
  Anti-T, Month 11 | 10.234 [9.128 to 11.475] | 11.004 [9.721 to 12.456] | 8.400 [7.285 to 9.685] | 13.016 [11.640 to 14.554]

19. Secondary Outcome: Number of Subjects With Anti-pertussis Toxoid (Anti-PT), Anti-filamentous Haemagglutinin (Anti-FHA) and Anti-pertactin (Anti-PRN) Concentrations ≥ the Cut-off Value
Description: The cut-off value for anti-PT, anti-FHA and anti-PRN concentrations was greater than or equal to (≥) 5 enzyme-linked immunosorbent assay (ELISA) units per milliliter (EL.U/mL).
Time Frame: Pre-primary vaccination at Month 0 and one month after final primary vaccination at Month 3
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix 3 Group | Nimenrix 2 Group | Menjugate Group | NeisVac-C Group
Number analyzed (Participants) | 117 | 112 | 123 | 115
Participants
  Anti-PT, Month 0: number analyzed (Participants) | 112 | 103 | 113 | 109
  Anti-PT, Month 0 | 23 | 32 | 28 | 31
  Anti-PT, Month 3: number analyzed (Participants) | 117 | 111 | 122 | 115
  Anti-PT, Month 3 | 117 | 111 | 122 | 115
  Anti-FHA, Month 0: number analyzed (Participants) | 114 | 104 | 115 | 109
  Anti-FHA, Month 0 | 83 | 85 | 93 | 78
  Anti-FHA, Month 3: number analyzed (Participants) | 117 | 111 | 123 | 115
  Anti-FHA, Month 3 | 117 | 111 | 123 | 115
  Anti-PRN, Month 0: number analyzed (Participants) | 115 | 104 | 116 | 110
  Anti-PRN, Month 0 | 31 | 39 | 44 | 32
  Anti-PRN, Month 3: number analyzed (Participants) | 117 | 112 | 122 | 115
  Anti-PRN, Month 3 | 117 | 112 | 122 | 115

20. Secondary Outcome: Anti-PT, Anti-FHA and Anti-PRN Antibody Concentrations
Description: Antibody concentrations were presented as geometric mean concentrations (GMCs) and expressed in EL.U/mL.
Time Frame: Pre-primary vaccination at Month 0 and one month after final primary vaccination at Month 3
Population: as for outcome 11
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Nimenrix 3 Group | Nimenrix 2 Group | Menjugate Group | NeisVac-C Group
Number analyzed (Participants) | 117 | 112 | 123 | 115
EL.U/mL
  Anti-PT, Month 0: number analyzed (Participants) | 112 | 103 | 113 | 109
  Anti-PT, Month 0 | 3.4 [3 to 3.8] | 3.9 [3.3 to 4.5] | 3.6 [3.2 to 4.2] | 4.1 [3.5 to 4.9]
  Anti-PT, Month 3: number analyzed (Participants) | 117 | 111 | 122 | 115
  Anti-PT, Month 3 | 52.7 [46.5 to 59.8] | 56.3 [49.5 to 64] | 56.5 [50.5 to 63.1] | 56.4 [50.6 to 63]
  Anti-FHA, Month 0: number analyzed (Participants) | 114 | 104 | 115 | 109
  Anti-FHA, Month 0 | 9.7 [8 to 11.9] | 13.2 [10.7 to 16.4] | 11.4 [9.4 to 13.9] | 11.9 [9.4 to 15.1]
  Anti-FHA, Month 3: number analyzed (Participants) | 117 | 111 | 123 | 115
  Anti-FHA, Month 3 | 124.3 [109 to 141.8] | 149.2 [131.2 to 169.6] | 139.1 [123.2 to 157.1] | 132 [115.1 to 151.3]
  Anti-PRN, Month 0: number analyzed (Participants) | 115 | 104 | 116 | 110
  Anti-PRN, Month 0 | 4 [3.4 to 4.7] | 5 [4 to 6.2] | 4.6 [3.9 to 5.4] | 4.7 [3.8 to 5.9]
  Anti-PRN, Month 3: number analyzed (Participants) | 117 | 112 | 122 | 115
  Anti-PRN, Month 3 | 122 [104.1 to 143.1] | 134.9 [119 to 152.9] | 118.2 [101.5 to 137.7] | 132 [113.6 to 153.5]

21. Secondary Outcome: Number of Subjects With Anti-PT, Anti-FHA and Anti-PRN Concentrations ≥ the Cut-off Value
Description: The cut-off value for anti-PT, anti-FHA and anti-PRN concentrations was greater than or equal to (≥) 5 EL.U/mL.
Time Frame: Pre-Booster dose at Month 10 and one month post-Booster dose at Month 11
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix 3 Group | Nimenrix 2 Group | Menjugate Group | NeisVac-C Group
Number analyzed (Participants) | 116 | 112 | 119 | 118
Participants
  Anti-PT, Month 10: number analyzed (Participants) | 114 | 112 | 118 | 116
  Anti-PT, Month 10 | 100 | 94 | 104 | 102
  Anti-PT, Month 11: number analyzed (Participants) | 110 | 109 | 116 | 116
  Anti-PT, Month 11 | 110 | 109 | 116 | 116
  Anti-FHA, Month 10: number analyzed (Participants) | 112 | 108 | 118 | 115
  Anti-FHA, Month 10 | 112 | 106 | 118 | 115
  Anti-FHA, Month 11: number analyzed (Participants) | 113 | 111 | 116 | 116
  Anti-FHA, Month 11 | 113 | 111 | 116 | 116
  Anti-PRN, Month 10: number analyzed (Participants) | 114 | 112 | 119 | 117
  Anti-PRN, Month 10 | 105 | 98 | 109 | 105
  Anti-PRN, Month 11: number analyzed (Participants) | 116 | 110 | 118 | 118
  Anti-PRN, Month 11 | 116 | 110 | 118 | 118

22. Secondary Outcome: Anti-PT, Anti-FHA and Anti-PRN Antibody Concentrations
Description: Antibody concentrations were presented as geometric mean concentrations (GMCs) and expressed in EL.U/mL.
Time Frame: Pre-Booster dose at Month 10 and one month post-Booster dose at Month 11
Population: as for outcome 13
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Nimenrix 3 Group | Nimenrix 2 Group | Menjugate Group | NeisVac-C Group
Number analyzed (Participants) | 116 | 112 | 119 | 118
EL.U/mL
  Anti-PT, Month 10: number analyzed (Participants) | 114 | 112 | 118 | 116
  Anti-PT, Month 10 | 11.0 [9.4 to 12.9] | 11.1 [9.4 to 13.1] | 13.1 [11.1 to 15.4] | 11.4 [9.9 to 13.3]
  Anti-PT, Month 11: number analyzed (Participants) | 110 | 109 | 116 | 116
  Anti-PT, Month 11 | 82.5 [71.9 to 94.7] | 78.2 [67.8 to 90.2] | 84.7 [73.5 to 97.5] | 82.7 [72.5 to 94.4]
  Anti-FHA, Month 10: number analyzed (Participants) | 112 | 108 | 118 | 115
  Anti-FHA, Month 10 | 34.5 [29.6 to 40.2] | 33.1 [27.5 to 39.8] | 37.4 [32.1 to 43.5] | 34.9 [29.8 to 40.9]
  Anti-FHA, Month 11: number analyzed (Participants) | 113 | 111 | 116 | 116
  Anti-FHA, Month 11 | 285.5 [250.6 to 325.4] | 296.3 [258.5 to 339.7] | 305.9 [269.0 to 347.8] | 302.9 [266.8 to 343.9]
  Anti-PRN, Month 10: number analyzed (Participants) | 114 | 112 | 119 | 117
  Anti-PRN, Month 10 | 17.9 [14.8 to 21.6] | 15.7 [13.1 to 18.8] | 19.9 [16.5 to 23.9] | 17.9 [14.8 to 21.6]
  Anti-PRN, Month 11: number analyzed (Participants) | 116 | 110 | 118 | 118
  Anti-PRN, Month 11 | 283.7 [233.9 to 344.1] | 290.8 [242.5 to 348.7] | 291.7 [246.1 to 345.7] | 334.3 [282.9 to 395.1]

23. Secondary Outcome: Number of Subjects With Anti-hepatitis B Surface Antigen (Anti-HBs) Antibody Concentrations Above the Cut-off Values
Description: The cut-off values for anti-HBs concentrations were greater than or equal to (≥) 10 milli-international units per milliliter (mIU/mL) and ≥ 100 mIU/mL.
Time Frame: Pre-primary vaccination at Month 0 and one month after final primary vaccination at Month 3
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix 3 Group | Nimenrix 2 Group | Menjugate Group | NeisVac-C Group
Number analyzed (Participants) | 98 | 84 | 97 | 93
Participants
  Anti-HBs ≥ 10 mIU/mL, Month 0: number analyzed (Participants) | 98 | 82 | 97 | 93
  Anti-HBs ≥ 10 mIU/mL, Month 0 | 33 | 34 | 39 | 28
  Anti-HBs ≥ 10 mIU/mL, Month 3: number analyzed (Participants) | 86 | 84 | 94 | 80
  Anti-HBs ≥ 10 mIU/mL, Month 3 | 85 | 84 | 94 | 79
  Anti-HBs ≥ 100 mIU/mL, Month 0: number analyzed (Participants) | 98 | 82 | 97 | 93
  Anti-HBs ≥ 100 mIU/mL, Month 0 | 17 | 14 | 14 | 8
  Anti-HBs ≥ 100 mIU/mL, Month 3: number analyzed (Participants) | 86 | 84 | 94 | 80
  Anti-HBs ≥ 100 mIU/mL, Month 3 | 74 | 79 | 89 | 73

24. Secondary Outcome: Anti-HBs Antibody Concentrations
Description: Antibody concentrations were presented as geometric mean concentrations (GMCs) and expressed in milli-international units per milliliter (mIU/mL).
Time Frame: Pre-primary vaccination at Month 0 and one month after final primary vaccination at Month 3
Population: as for outcome 11
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | Nimenrix 3 Group | Nimenrix 2 Group | Menjugate Group | NeisVac-C Group
Number analyzed (Participants) | 98 | 84 | 97 | 93
mIU/mL
  Anti-HBs, Month 0: number analyzed (Participants) | 98 | 82 | 97 | 93
  Anti-HBs, Month 0 | 12.0 [7.6 to 18.7] | 13.7 [8.4 to 22.4] | 11.3 [7.7 to 16.7] | 7.5 [5.4 to 10.5]
  Anti-HBs, Month 3: number analyzed (Participants) | 86 | 84 | 94 | 80
  Anti-HBs, Month 3 | 692.3 [513.2 to 934.0] | 732.2 [555.1 to 965.8] | 848.3 [663.7 to 1084.1] | 729.5 [530.3 to 1003.5]

25. Secondary Outcome: Number of Subjects With Anti-HBs Antibody Concentrations Above the Cut-off Values
Description: The cut-off values for anti-HBs concentrations were greater than or equal to (≥) 10 mIU/mL and ≥ 100 mIU/mL.
Time Frame: Pre-Booster dose at Month 10 and one month post-Booster dose at Month 11
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix 3 Group | Nimenrix 2 Group | Menjugate Group | NeisVac-C Group
Number analyzed (Participants) | 98 | 97 | 103 | 100
Participants
  Anti-HBs ≥ 10 mIU/mL, Month 10: number analyzed (Participants) | 98 | 91 | 101 | 100
  Anti-HBs ≥ 10 mIU/mL, Month 10 | 91 | 86 | 96 | 94
  Anti-HBs ≥ 10 mIU/mL, Month 11: number analyzed (Participants) | 97 | 97 | 103 | 100
  Anti-HBs ≥ 10 mIU/mL, Month 11 | 95 | 97 | 103 | 100
  Anti-HBs ≥ 100 mIU/mL, Month 10: number analyzed (Participants) | 98 | 91 | 101 | 100
  Anti-HBs ≥ 100 mIU/mL, Month 10 | 67 | 58 | 75 | 65
  Anti-HBs ≥ 100 mIU/mL, Month 11: number analyzed (Participants) | 97 | 97 | 103 | 100
  Anti-HBs ≥ 100 mIU/mL, Month 11 | 93 | 97 | 102 | 97

26. Secondary Outcome: Anti-HBs Antibody Concentrations
Description: as for outcome 24
Time Frame: Pre-Booster dose at Month 10 and one month post-Booster dose at Month 11
Population: as for outcome 13
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | Nimenrix 3 Group | Nimenrix 2 Group | Menjugate Group | NeisVac-C Group
Number analyzed (Participants) | 98 | 97 | 103 | 100
mIU/mL
  Anti-HBs, Month 10: number analyzed (Participants) | 98 | 91 | 101 | 100
  Anti-HBs, Month 10 | 150.5 [111.4 to 203.3] | 138.2 [99.3 to 192.3] | 196.6 [141.6 to 273.1] | 141.9 [106.5 to 189.0]
  Anti-HBs, Month 11: number analyzed (Participants) | 97 | 97 | 103 | 100
  Anti-HBs, Month 11 | 3624.9 [2570.0 to 5112.8] | 4129.8 [3095.4 to 5509.8] | 4866.4 [3723.5 to 6360.1] | 3878.7 [2861.7 to 5257.3]

27. Secondary Outcome: Number of Subjects With Anti-polyribosyl Ribitol Phosphate (Anti-PRP) Concentrations ≥ the Cut-off Values
Description: The cut-off values for anti-PRP antibody concentrations were greater than or equal to (≥) 0.15 micrograms per milliliter (µg/mL) and ≥ 1.0 µg/mL.
Time Frame: Pre-primary vaccination at Month 0 and one month after final primary vaccination at Month 3
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix 3 Group | Nimenrix 2 Group | Menjugate Group | NeisVac-C Group
Number analyzed (Participants) | 119 | 113 | 123 | 114
Participants
  Anti-PRP ≥ 0.15 µg/mL, Month 0: number analyzed (Participants) | 113 | 106 | 113 | 109
  Anti-PRP ≥ 0.15 µg/mL, Month 0 | 46 | 55 | 46 | 47
  Anti-PRP ≥ 0.15 µg/mL, Month 3 | 119 | 113 | 121 | 113
  Anti-PRP ≥ 1.0 µg/mL, Month 0: number analyzed (Participants) | 113 | 106 | 113 | 109
  Anti-PRP ≥ 1.0 µg/mL, Month 0 | 9 | 19 | 10 | 7
  Anti-PRP ≥ 1.0 µg/mL, Month 3 | 106 | 101 | 94 | 106

28. Secondary Outcome: Anti-PRP Antibody Concentrations
Description: Antibody concentrations were presented as geometric mean concentrations (GMCs) and expressed in micrograms per milliliter (µg/mL).
Time Frame: Pre-primary vaccination at Month 0 and one month after final primary vaccination at Month 3
Population: as for outcome 11
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | Nimenrix 3 Group | Nimenrix 2 Group | Menjugate Group | NeisVac-C Group
Number analyzed (Participants) | 119 | 113 | 123 | 114
µg/mL
  Anti-PRP, Month 0 | 0.158 [0.131 to 0.191] | 0.213 [0.168 to 0.27] | 0.162 [0.132 to 0.198] | 0.162 [0.133 to 0.196]
  Anti-PRP, Month 3 | 4.011 [3.275 to 4.912] | 3.573 [2.946 to 4.334] | 2.752 [2.144 to 3.534] | 4.662 [3.788 to 5.739]

29. Secondary Outcome: Number of Subjects With Anti-PRP Antibody Concentrations Above the Cut-off Values
Description: The cut-off values for anti-PRP antibody concentrations were greater than or equal to (≥) 0.15 µg/mL and ≥ 1.0 µg/mL.
Time Frame: Pre-Booster dose at Month 10 and one month post-Booster dose at Month 11
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix 3 Group | Nimenrix 2 Group | Menjugate Group | NeisVac-C Group
Number analyzed (Participants) | 116 | 112 | 119 | 118
Participants
  Anti-PRP ≥ 0.15 µg/mL, Month 10: number analyzed (Participants) | 114 | 112 | 119 | 117
  Anti-PRP ≥ 0.15 µg/mL, Month 10 | 92 | 91 | 91 | 100
  Anti-PRP ≥ 0.15 µg/mL, Month 11 | 116 | 112 | 119 | 118
  Anti-PRP ≥ 1.0 µg/mL, Month 10: number analyzed (Participants) | 114 | 112 | 119 | 117
  Anti-PRP ≥ 1.0 µg/mL, Month 10 | 23 | 20 | 40 | 31
  Anti-PRP ≥ 1.0 µg/mL, Month 11 | 113 | 112 | 119 | 114

30. Secondary Outcome: Anti-PRP Antibody Concentrations
Description: as for outcome 28
Time Frame: Pre-Booster dose at Month 10 and one month post-Booster dose at Month 11
Population: as for outcome 13
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | Nimenrix 3 Group | Nimenrix 2 Group | Menjugate Group | NeisVac-C Group
Number analyzed (Participants) | 116 | 112 | 119 | 118
µg/mL
  Anti-PRP, Month 10: number analyzed (Participants) | 114 | 112 | 119 | 117
  Anti-PRP, Month 10 | 0.378 [0.308 to 0.464] | 0.400 [0.324 to 0.494] | 0.535 [0.404 to 0.707] | 0.535 [0.427 to 0.671]
  Anti-PRP, Month 11 | 17.350 [14.124 to 21.313] | 17.519 [14.041 to 21.859] | 22.879 [18.147 to 28.847] | 23.973 [19.194 to 29.941]

31. Secondary Outcome: Number of Subjects With Anti-poliovirus Type 1, 2 and 3 Antibody Concentrations ≥ the Cut-off Value
Description: The cut-off value for anti-poliovirus type 1, 2 and 3 antibody concentrations was greater than or equal to (≥) 1:8.
Time Frame: Pre-primary vaccination at Month 0 and one month after final primary vaccination at Month 3
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix 3 Group | Nimenrix 2 Group | Menjugate Group | NeisVac-C Group
Number analyzed (Participants) | 93 | 83 | 90 | 86
Participants
  Anti-Polio 1, Month 0: number analyzed (Participants) | 71 | 58 | 72 | 58
  Anti-Polio 1, Month 0 | 52 | 46 | 54 | 46
  Anti-Polio 1, Month 3: number analyzed (Participants) | 91 | 83 | 90 | 86
  Anti-Polio 1, Month 3 | 91 | 83 | 89 | 84
  Anti-Polio 2, Month 0: number analyzed (Participants) | 64 | 54 | 66 | 62
  Anti-Polio 2, Month 0 | 39 | 40 | 44 | 41
  Anti-Polio 2, Month 3: number analyzed (Participants) | 81 | 71 | 81 | 72
  Anti-Polio 2, Month 3 | 81 | 70 | 81 | 70
  Anti-Polio 3, Month 0: number analyzed (Participants) | 58 | 52 | 60 | 51
  Anti-Polio 3, Month 0 | 21 | 21 | 11 | 23
  Anti-Polio 3, Month 3: number analyzed (Participants) | 93 | 79 | 87 | 78
  Anti-Polio 3, Month 3 | 93 | 79 | 87 | 77

32. Secondary Outcome: Anti-polio Type 1, 2 and 3 Antibody Titers
Description: Antibody titers were presented as geometric mean titers (GMTs).
Time Frame: Pre-primary vaccination at Month 0 and one month after final primary vaccination at Month 3
Population: as for outcome 11
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Nimenrix 3 Group | Nimenrix 2 Group | Menjugate Group | NeisVac-C Group
Number analyzed (Participants) | 93 | 83 | 90 | 86
Titers
  Anti-Polio 1, Month 0: number analyzed (Participants) | 71 | 58 | 72 | 58
  Anti-Polio 1, Month 0 | 32.7 [22.5 to 47.5] | 40.2 [27.3 to 59.3] | 28.1 [20.1 to 39.3] | 30.7 [21.5 to 43.9]
  Anti-Polio 1, Month 3: number analyzed (Participants) | 91 | 83 | 90 | 86
  Anti-Polio 1, Month 3 | 279.6 [222.4 to 351.5] | 317.9 [227.6 to 444] | 424.1 [323.1 to 556.6] | 277.7 [200.7 to 384.1]
  Anti-Polio 2, Month 0: number analyzed (Participants) | 64 | 54 | 66 | 62
  Anti-Polio 2, Month 0 | 19.4 [13.2 to 28.7] | 28 [18.4 to 42.5] | 17.4 [12.7 to 23.8] | 22.9 [15.6 to 33.5]
  Anti-Polio 2, Month 3: number analyzed (Participants) | 81 | 71 | 81 | 72
  Anti-Polio 2, Month 3 | 225.2 [173.2 to 292.6] | 244.8 [173.3 to 345.9] | 274.5 [202.1 to 372.8] | 232.7 [160.8 to 336.6]
  Anti-Polio 3, Month 0: number analyzed (Participants) | 58 | 52 | 60 | 51
  Anti-Polio 3, Month 0 | 11.5 [7.6 to 17.5] | 11.7 [7.8 to 17.5] | 5.9 [4.7 to 7.5] | 14.2 [8.8 to 22.8]
  Anti-Polio 3, Month 3: number analyzed (Participants) | 93 | 79 | 87 | 78
  Anti-Polio 3, Month 3 | 642.7 [478.7 to 862.8] | 675 [486.3 to 936.9] | 674 [525.5 to 864.5] | 494.3 [347.4 to 703.3]

33. Secondary Outcome: Number of Subjects With Anti-polio Type 1, 2 and 3 Antibody Concentrations ≥ the Cut-off Value
Description: The cut-off value for anti-poliovirus type 1, 2 and 3 antibody concentrations was greater than or equal to (≥) 1:8.
Time Frame: Pre-Booster dose at Month 10 and one month post-Booster dose at Month 11
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix 3 Group | Nimenrix 2 Group | Menjugate Group | NeisVac-C Group
Number analyzed (Participants) | 85 | 85 | 86 | 87
Participants
  Anti-Polio 1, Month 10: number analyzed (Participants) | 80 | 68 | 82 | 87
  Anti-Polio 1, Month 10 | 74 | 63 | 80 | 81
  Anti-Polio 1, Month 11: number analyzed (Participants) | 85 | 85 | 81 | 84
  Anti-Polio 1, Month 11 | 85 | 85 | 81 | 84
  Anti-Polio 2, Month 10: number analyzed (Participants) | 71 | 70 | 86 | 77
  Anti-Polio 2, Month 10 | 69 | 66 | 83 | 72
  Anti-Polio 2, Month 11: number analyzed (Participants) | 70 | 74 | 71 | 68
  Anti-Polio 2, Month 11 | 70 | 74 | 71 | 68
  Anti-Polio 3, Month 10: number analyzed (Participants) | 61 | 65 | 63 | 68
  Anti-Polio 3, Month 10 | 57 | 62 | 62 | 64
  Anti-Polio 3, Month 11: number analyzed (Participants) | 79 | 67 | 74 | 69
  Anti-Polio 3, Month 11 | 79 | 67 | 74 | 69

34. Secondary Outcome: Anti-polio Type 1, 2 and 3 Antibody Titers
Description: Antibody titers were presented as geometric mean titers (GMTs).
Time Frame: Pre-Booster dose at Month 10 and one month post-Booster dose at Month 11
Population: as for outcome 13
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Nimenrix 3 Group | Nimenrix 2 Group | Menjugate Group | NeisVac-C Group
Number analyzed (Participants) | 85 | 85 | 86 | 87
Titers
  Anti-polio 1, Month 10: number analyzed (Participants) | 80 | 68 | 82 | 87
  Anti-polio 1, Month 10 | 74.9 [56.3 to 99.6] | 84.7 [60.0 to 119.7] | 120.8 [92.5 to 157.8] | 90.0 [65.8 to 123.0]
  Anti-polio 1, Month 11: number analyzed (Participants) | 85 | 85 | 81 | 84
  Anti-polio 1, Month 11 | 909.8 [694.1 to 1192.6] | 1070.9 [812.5 to 1411.4] | 1524.5 [1214.9 to 1913.0] | 1217.7 [956.5 to 1550.2]
  Anti-polio 2, Month 10: number analyzed (Participants) | 71 | 70 | 86 | 77
  Anti-polio 2, Month 10 | 93.7 [71.1 to 123.5] | 80.1 [57.6 to 111.5] | 112.5 [86.7 to 146.1] | 78.1 [57.6 to 105.9]
  Anti-polio 2, Month 11: number analyzed (Participants) | 70 | 74 | 71 | 68
  Anti-polio 2, Month 11 | 1205.7 [902.2 to 1611.3] | 1306.3 [985.1 to 1732.2] | 2068.0 [1602.7 to 2668.5] | 1419.0 [1088.4 to 1849.9]
  Anti-polio 3, Month 10: number analyzed (Participants) | 61 | 65 | 63 | 68
  Anti-polio 3, Month 10 | 115.0 [80.1 to 165.2] | 104.6 [77.9 to 140.3] | 155.2 [118.3 to 203.7] | 108.6 [77.6 to 152.1]
  Anti-polio 3, Month 11: number analyzed (Participants) | 79 | 67 | 74 | 69
  Anti-polio 3, Month 11 | 1681.0 [1285.1 to 2198.9] | 2167.8 [1645.7 to 2855.6] | 2136.2 [1688.1 to 2703.4] | 1852.2 [1425.6 to 2406.4]

35. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms
Description: Assessed solicited local symptoms were pain, redness and swelling. Any = occurrence of the symptom regardless of intensity grade. Grade 3 pain = cried when limb was moved/spontaneously painful. Grade 3 redness/swelling = redness/swelling spreading beyond 30 millimeters (mm) of injection site. For the Nimenrix 2, Menjugate and NeisVac-C groups, results corresponding to Dose 2 are for Infanrix hexa and Synflorix vaccination at Visit 2 (Month 1), while results corresponding to Dose 3 refer to the vaccination at Visit 3 (Month 2).
Time Frame: During the 8-day (Days 0-7) post-vaccination period following each dose and across doses from Day 0 to Month 3 (Primary Vaccination)
Population: The analysis was performed on the Primary Total Vaccinated cohort, which included all vaccinated subjects during the primary phase, who had filled in their symptom sheets. For the considered assay and time point data was reported only for the Primary Vaccination doses.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix 3 Group | Nimenrix 2 Group | Menjugate Group | NeisVac-C Group
Number analyzed (Participants) | 518 | 523 | 509 | 518
Participants
  Any Pain, Dose 1: number analyzed (Participants) | 518 | 523 | 509 | 517
  Any Pain, Dose 1 | 247 | 243 | 243 | 233
  Grade 3 Pain, Dose 1: number analyzed (Participants) | 518 | 523 | 509 | 517
  Grade 3 Pain, Dose 1 | 32 | 33 | 28 | 34
  Any Redness, Dose 1: number analyzed (Participants) | 518 | 523 | 509 | 517
  Any Redness, Dose 1 | 241 | 229 | 236 | 230
  Grade 3 Redness, Dose 1: number analyzed (Participants) | 518 | 523 | 509 | 517
  Grade 3 Redness, Dose 1 | 9 | 5 | 9 | 5
  Any Swelling, Dose 1: number analyzed (Participants) | 518 | 523 | 509 | 517
  Any Swelling, Dose 1 | 188 | 182 | 179 | 188
  Grade 3 Swelling, Dose 1: number analyzed (Participants) | 518 | 523 | 509 | 517
  Grade 3 Swelling, Dose 1 | 6 | 4 | 14 | 6
  Any Pain, Dose 2: number analyzed (Participants) | 511 | 517 | 509 | 513
  Any Pain, Dose 2 | 212 | 210 | 230 | 214
  Grade 3 Pain, Dose 2: number analyzed (Participants) | 511 | 517 | 509 | 513
  Grade 3 Pain, Dose 2 | 23 | 37 | 23 | 29
  Any Redness, Dose 2: number analyzed (Participants) | 511 | 517 | 509 | 513
  Any Redness, Dose 2 | 261 | 271 | 283 | 284
  Grade 3 Redness, Dose 2: number analyzed (Participants) | 511 | 517 | 509 | 513
  Grade 3 Redness, Dose 2 | 3 | 5 | 10 | 2
  Any Swelling, Dose 2: number analyzed (Participants) | 511 | 517 | 509 | 513
  Any Swelling, Dose 2 | 211 | 206 | 225 | 210
  Grade 3 Swelling, Dose 2: number analyzed (Participants) | 511 | 517 | 509 | 513
  Grade 3 Swelling, Dose 2 | 3 | 6 | 14 | 10
  Any Pain, Dose 3: number analyzed (Participants) | 505 | 517 | 507 | 508
  Any Pain, Dose 3 | 168 | 180 | 180 | 193
  Grade 3 Pain, Dose 3: number analyzed (Participants) | 505 | 517 | 507 | 508
  Grade 3 Pain, Dose 3 | 13 | 18 | 15 | 22
  Any Redness, Dose 3: number analyzed (Participants) | 505 | 517 | 507 | 508
  Any Redness, Dose 3 | 247 | 265 | 308 | 274
  Grade 3 Redness, Dose 3: number analyzed (Participants) | 505 | 517 | 507 | 508
  Grade 3 Redness, Dose 3 | 9 | 6 | 13 | 9
  Any Swelling, Dose 3: number analyzed (Participants) | 505 | 517 | 507 | 508
  Any Swelling, Dose 3 | 210 | 216 | 252 | 218
  Grade 3 Swelling, Dose 3: number analyzed (Participants) | 505 | 517 | 507 | 508
  Grade 3 Swelling, Dose 3 | 8 | 6 | 11 | 13
  Any Pain, Across doses | 319 | 332 | 344 | 327
  Grade 3 Pain, Across doses | 54 | 67 | 48 | 69
  Any Redness, Across doses | 363 | 369 | 391 | 371
  Grade 3 Redness, Across doses | 18 | 15 | 24 | 15
  Any Swelling, Across doses | 326 | 318 | 343 | 317
  Grade 3 Swelling, Across doses | 15 | 11 | 27 | 24

36. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms Post-meningococcal Vaccination
Description: Assessed solicited local symptoms were pain, redness and swelling. Any = occurrence of the symptom regardless of intensity grade. Grade 3 pain = cried when limb was moved/spontaneously painful. Grade 3 redness/swelling = redness/swelling spreading beyond 30 millimeters (mm) of injection site.
Time Frame: During the 8-day (Days 0-7) post-meningococcal vaccination period following each dose and across doses from Day 0 to Month 3 (Primary Vaccination)
Population: The analysis was performed on the Primary Total Vaccinated cohort, which included all vaccinated subjects during the primary phase, who had filled in their symptom sheets. No data was applicable for the Nimenrix 2 Group, Menjugate Group and NeisVac-C Group since meningococcal vaccine was not given in Dose 2.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix 3 Group | Nimenrix 2 Group | Menjugate Group | NeisVac-C Group
Number analyzed (Participants) | 518 | 523 | 509 | 518
Participants
  Any Pain, Dose 1: number analyzed (Participants) | 518 | 523 | 509 | 517
  Any Pain, Dose 1 | 161 | 155 | 158 | 157
  Grade 3 Pain, Dose 1: number analyzed (Participants) | 518 | 523 | 509 | 517
  Grade 3 Pain, Dose 1 | 18 | 17 | 12 | 24
  Any Redness, Dose 1: number analyzed (Participants) | 518 | 523 | 509 | 517
  Any Redness, Dose 1 | 132 | 128 | 138 | 140
  Grade 3 Redness, Dose 1: number analyzed (Participants) | 518 | 523 | 509 | 517
  Grade 3 Redness, Dose 1 | 2 | 1 | 2 | 1
  Any Swelling, Dose 1: number analyzed (Participants) | 518 | 523 | 509 | 517
  Any Swelling, Dose 1 | 68 | 62 | 87 | 82
  Grade 3 Swelling, Dose 1: number analyzed (Participants) | 518 | 523 | 509 | 517
  Grade 3 Swelling, Dose 1 | 1 | 0 | 3 | 0
  Any Pain, Dose 2: number analyzed (Participants) | 510 | 0 | 0 | 0
  Any Pain, Dose 2 | 125 | 0 | 0 | 0
  Grade 3 Pain, Dose 2: number analyzed (Participants) | 510 | 0 | 0 | 0
  Grade 3 Pain, Dose 2 | 9 | 0 | 0 | 0
  Any Redness, Dose 2: number analyzed (Participants) | 510 | 0 | 0 | 0
  Any Redness, Dose 2 | 131 | 0 | 0 | 0
  Grade 3 Redness, Dose 2: number analyzed (Participants) | 510 | 0 | 0 | 0
  Grade 3 Redness, Dose 2 | 0 | 0 | 0 | 0
  Any Swelling, Dose 2: number analyzed (Participants) | 510 | 0 | 0 | 0
  Any Swelling, Dose 2 | 77 | 0 | 0 | 0
  Grade 3 Swelling, Dose 2: number analyzed (Participants) | 510 | 0 | 0 | 0
  Grade 3 Swelling, Dose 2 | 0 | 0 | 0 | 0
  Any Pain, Dose 3: number analyzed (Participants) | 505 | 516 | 507 | 507
  Any Pain, Dose 3 | 106 | 124 | 130 | 142
  Grade 3 Pain, Dose 3: number analyzed (Participants) | 505 | 516 | 507 | 507
  Grade 3 Pain, Dose 3 | 7 | 11 | 9 | 12
  Any Redness, Dose 3: number analyzed (Participants) | 505 | 516 | 507 | 507
  Any Redness, Dose 3 | 162 | 169 | 214 | 197
  Grade 3 Redness, Dose 3: number analyzed (Participants) | 505 | 516 | 507 | 507
  Grade 3 Redness, Dose 3 | 0 | 0 | 0 | 1
  Any Swelling, Dose 3: number analyzed (Participants) | 505 | 516 | 507 | 507
  Any Swelling, Dose 3 | 104 | 115 | 137 | 130
  Grade 3 Swelling, Dose 3: number analyzed (Participants) | 505 | 516 | 507 | 507
  Grade 3 Swelling, Dose 3 | 0 | 1 | 0 | 4
  Any Pain, Across doses | 229 | 202 | 213 | 212
  Grade 3 Pain, Across doses | 29 | 26 | 19 | 33
  Any Redness, Across doses | 233 | 206 | 255 | 233
  Grade 3 Redness, Across doses | 2 | 1 | 2 | 2
  Any Swelling, Across doses | 154 | 136 | 175 | 164
  Grade 3 Swelling, Across doses | 1 | 1 | 3 | 4

37. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms Post-Infanrix™ Hexa Vaccination
Description: as for outcome 36
Time Frame: During the 8-day (Days 0-7) post-Infanrix hexa vaccination period following each dose and across doses from Day 0 to Month 3 (Primary Vaccination)
Population: as for outcome 35
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix 3 Group | Nimenrix 2 Group | Menjugate Group | NeisVac-C Group
Number analyzed (Participants) | 518 | 523 | 509 | 518
Participants
  Any Pain, Dose 1: number analyzed (Participants) | 518 | 523 | 509 | 517
  Any Pain, Dose 1 | 212 | 202 | 208 | 210
  Grade 3 Pain, Dose 1: number analyzed (Participants) | 518 | 523 | 509 | 517
  Grade 3 Pain, Dose 1 | 28 | 28 | 25 | 32
  Any Redness, Dose 1: number analyzed (Participants) | 518 | 523 | 509 | 517
  Any Redness, Dose 1 | 201 | 190 | 191 | 192
  Grade 3 Redness, Dose 1: number analyzed (Participants) | 518 | 523 | 509 | 517
  Grade 3 Redness, Dose 1 | 7 | 3 | 6 | 2
  Any Swelling, Dose 1: number analyzed (Participants) | 518 | 523 | 509 | 517
  Any Swelling, Dose 1 | 148 | 148 | 128 | 147
  Grade 3 Swelling, Dose 1 | 6 | 4 | 13 | 4
  Any Pain, Dose 2: number analyzed (Participants) | 511 | 517 | 509 | 513
  Any Pain, Dose 2 | 184 | 200 | 219 | 198
  Grade 3 Pain, Dose 2: number analyzed (Participants) | 511 | 517 | 509 | 513
  Grade 3 Pain, Dose 2 | 18 | 34 | 22 | 27
  Any Redness, Dose 2: number analyzed (Participants) | 511 | 517 | 509 | 513
  Any Redness, Dose 2 | 232 | 250 | 264 | 265
  Grade 3 Redness, Dose 2: number analyzed (Participants) | 511 | 517 | 509 | 513
  Grade 3 Redness, Dose 2 | 1 | 5 | 10 | 2
  Any Swelling, Dose 2: number analyzed (Participants) | 511 | 517 | 509 | 513
  Any Swelling, Dose 2 | 182 | 185 | 208 | 195
  Grade 3 Swelling, Dose 2: number analyzed (Participants) | 511 | 517 | 509 | 513
  Grade 3 Swelling, Dose 2 | 1 | 3 | 13 | 10
  Any Pain, Dose 3: number analyzed (Participants) | 505 | 517 | 507 | 508
  Any Pain, Dose 3 | 144 | 159 | 153 | 175
  Grade 3 Pain, Dose 3: number analyzed (Participants) | 505 | 517 | 507 | 508
  Grade 3 Pain, Dose 3 | 9 | 14 | 11 | 19
  Any Redness, Dose 3: number analyzed (Participants) | 505 | 517 | 507 | 508
  Any Redness, Dose 3 | 228 | 243 | 272 | 247
  Grade 3 Redness, Dose 3: number analyzed (Participants) | 505 | 517 | 507 | 508
  Grade 3 Redness, Dose 3 | 5 | 4 | 11 | 7
  Any Swelling, Dose 3: number analyzed (Participants) | 505 | 517 | 507 | 508
  Any Swelling, Dose 3 | 191 | 200 | 227 | 197
  Grade 3 Swelling, Dose 3: number analyzed (Participants) | 505 | 517 | 507 | 508
  Grade 3 Swelling, Dose 3 | 6 | 4 | 11 | 11
  Any Pain, Across doses | 289 | 311 | 314 | 310
  Grade 3 Pain, Across doses | 44 | 58 | 43 | 63
  Any Redness, Across doses | 336 | 344 | 358 | 349
  Grade 3 Redness, Across doses | 13 | 11 | 19 | 10
  Any Swelling, Across doses | 297 | 292 | 308 | 294
  Grade 3 Swelling, Across doses | 12 | 7 | 25 | 21

38. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms Post-Synflorix Vaccination
Description: as for outcome 36
Time Frame: During the 8-day (Days 0-7) post-Synflorix vaccination period following each dose and across doses from Day 0 to Month 3 (Primary Vaccination)
Population: as for outcome 35
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix 3 Group | Nimenrix 2 Group | Menjugate Group | NeisVac-C Group
Number analyzed (Participants) | 518 | 523 | 509 | 518
Participants
  Any Pain, Dose 1: number analyzed (Participants) | 518 | 523 | 509 | 517
  Any Pain, Dose 1 | 218 | 201 | 217 | 195
  Grade 3 Pain, Dose 1: number analyzed (Participants) | 518 | 523 | 509 | 517
  Grade 3 Pain, Dose 1 | 29 | 26 | 26 | 32
  Any Redness, Dose 1: number analyzed (Participants) | 518 | 523 | 509 | 517
  Any Redness, Dose 1 | 209 | 184 | 196 | 183
  Grade 3 Redness, Dose 1: number analyzed (Participants) | 518 | 523 | 509 | 517
  Grade 3 Redness, Dose 1 | 4 | 2 | 5 | 4
  Any Swelling, Dose 1: number analyzed (Participants) | 518 | 523 | 509 | 517
  Any Swelling, Dose 1 | 135 | 136 | 130 | 120
  Grade 3 Swelling, Dose 1: number analyzed (Participants) | 518 | 523 | 509 | 517
  Grade 3 Swelling, Dose 1 | 4 | 1 | 10 | 4
  Any Pain, Dose 2: number analyzed (Participants) | 511 | 517 | 509 | 513
  Any Pain, Dose 2 | 179 | 186 | 203 | 189
  Grade 3 Pain, Dose 2: number analyzed (Participants) | 511 | 517 | 509 | 513
  Grade 3 Pain, Dose 2 | 20 | 31 | 19 | 25
  Any Redness, Dose 2: number analyzed (Participants) | 511 | 517 | 509 | 513
  Any Redness, Dose 2 | 197 | 216 | 225 | 235
  Grade 3 Redness, Dose 2: number analyzed (Participants) | 511 | 517 | 509 | 513
  Grade 3 Redness, Dose 2 | 2 | 1 | 5 | 1
  Any Swelling, Dose 2: number analyzed (Participants) | 511 | 517 | 509 | 513
  Any Swelling, Dose 2 | 154 | 162 | 156 | 155
  Grade 3 Swelling, Dose 2: number analyzed (Participants) | 511 | 517 | 509 | 513
  Grade 3 Swelling, Dose 2 | 3 | 4 | 8 | 5
  Any Pain, Dose 3: number analyzed (Participants) | 505 | 517 | 507 | 508
  Any Pain, Dose 3 | 129 | 152 | 132 | 150
  Grade 3 Pain, Dose 3: number analyzed (Participants) | 505 | 517 | 507 | 508
  Grade 3 Pain, Dose 3 | 10 | 13 | 10 | 18
  Any Redness, Dose 3: number analyzed (Participants) | 505 | 517 | 507 | 508
  Any Redness, Dose 3 | 173 | 213 | 227 | 209
  Grade 3 Redness, Dose 3: number analyzed (Participants) | 505 | 517 | 507 | 508
  Grade 3 Redness, Dose 3 | 4 | 4 | 6 | 2
  Any Swelling, Dose 3: number analyzed (Participants) | 505 | 517 | 507 | 508
  Any Swelling, Dose 3 | 136 | 152 | 164 | 146
  Grade 3 Swelling, Dose 3: number analyzed (Participants) | 505 | 517 | 507 | 508
  Grade 3 Swelling, Dose 3 | 3 | 4 | 6 | 5
  Any Pain, Across doses | 285 | 304 | 312 | 291
  Grade 3 Pain, Across doses | 46 | 54 | 41 | 61
  Any Redness, Across doses | 297 | 322 | 331 | 316
  Grade 3 Redness, Across doses | 8 | 7 | 12 | 7
  Any Swelling, Across doses | 247 | 259 | 262 | 237
  Grade 3 Swelling, Across doses | 9 | 7 | 16 | 13

39. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms Post-meningococcal Vaccination
Description: as for outcome 36
Time Frame: During the 8-day (Days 0-7) post-meningococcal booster vaccination period
Population: The analysis was performed on the Booster Total Vaccinated cohort, which included all vaccinated subjects during the booster phase, who had filled in their symptom sheets.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix 3 Group | Nimenrix 2 Group | Menjugate Group | NeisVac-C Group
Number analyzed (Participants) | 491 | 510 | 496 | 503
Participants
  Any Pain | 191 | 203 | 203 | 181
  Grade 3 Pain | 24 | 23 | 31 | 18
  Any Redness | 186 | 221 | 213 | 228
  Grade 3 Redness | 3 | 6 | 5 | 4
  Any Swelling | 133 | 152 | 158 | 165
  Grade 3 Swelling | 1 | 2 | 2 | 5

40. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms Post-Infanrix™ Hexa Vaccination
Description: as for outcome 36
Time Frame: During the 8-day (Days 0-7) post-Infanrix™ hexa booster vaccination period
Population: as for outcome 39
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix 3 Group | Nimenrix 2 Group | Menjugate Group | NeisVac-C Group
Number analyzed (Participants) | 491 | 510 | 495 | 504
Participants
  Any Pain | 240 | 241 | 242 | 221
  Grade Pain | 35 | 33 | 39 | 23
  Any Redness | 259 | 286 | 282 | 280
  Grade 3 Redness | 29 | 24 | 32 | 22
  Any Swelling | 212 | 226 | 244 | 240
  Grade 3 Swelling | 20 | 18 | 17 | 14

41. Secondary Outcome: Number of Subjects With Any Unsolicited Adverse Events (AEs)
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination.
Time Frame: Within 31-days (Days 0-30) post-each primary vaccination dose
Population: The analysis was performed on the Primary Total Vaccinated cohort, which included all vaccinated subjects during the primary phase, who had filled in their symptom sheets.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix 3 Group | Nimenrix 2 Group | Menjugate Group | NeisVac-C Group
Number analyzed (Participants) | 528 | 524 | 516 | 527
Participants | 293 | 273 | 291 | 280

42. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms Post-Synflorix™ Vaccination
Description: as for outcome 36
Time Frame: During the 8-day (Days 0-7) post-Synflorix™ booster vaccination period
Population: as for outcome 39
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix 3 Group | Nimenrix 2 Group | Menjugate Group | NeisVac-C Group
Number analyzed (Participants) | 491 | 510 | 495 | 504
Participants
  Any Pain | 212 | 215 | 227 | 205
  Grade 3 Pain | 36 | 33 | 33 | 26
  Any Redness | 219 | 243 | 242 | 250
  Grade 3 Redness | 14 | 9 | 20 | 9
  Any Swelling | 173 | 174 | 189 | 193
  Grade 3 Swelling | 5 | 5 | 4 | 10

43. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms
Description: Assessed solicited general symptoms were drowsiness, irritability, loss of appetite and temperature [defined as rectal temperature greater than or equal to (≥) 38 degrees Celsius (°C)]. Any = occurrence of any general symptoms, regardless of their intensity grade or relationship to study vaccination. Grade 3 Drowsiness = Drowsiness that prevented normal activity. Grade 3 Irritability = Crying that could not be comforted/prevented normal activity. Grade 3 Loss of appetite = Not eating at all. Grade 3 Temperature= temperature above 40.0 (°C). Related = symptom assessed by the investigator as related to the vaccination. For the Nimenrix 2, Menjugate and NeisVac-C groups, results corresponding to Dose 2 are for Infanrix™ hexa and Synflorix™ vaccination at Visit 2 (Month 1), while results corresponding to Dose 3 refer to the vaccination at Visit 3 (Month 2).
Time Frame: as for outcome 35
Population: as for outcome 41
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix 3 Group | Nimenrix 2 Group | Menjugate Group | NeisVac-C Group
Number analyzed (Participants) | 518 | 523 | 509 | 518
Participants
  Any Drowsiness, Dose 1: number analyzed (Participants) | 518 | 523 | 508 | 517
  Any Drowsiness, Dose 1 | 298 | 282 | 285 | 297
  Grade 3 Drowsiness, Dose 1: number analyzed (Participants) | 518 | 523 | 508 | 517
  Grade 3 Drowsiness, Dose 1 | 22 | 22 | 17 | 34
  Related Drowsiness, Dose 1: number analyzed (Participants) | 518 | 523 | 508 | 517
  Related Drowsiness, Dose 1 | 163 | 167 | 163 | 178
  Any Irritability, Dose 1: number analyzed (Participants) | 518 | 523 | 508 | 517
  Any Irritability, Dose 1 | 329 | 337 | 355 | 364
  Grade 3 Irritability, Dose 1: number analyzed (Participants) | 518 | 523 | 508 | 517
  Grade 3 Irritability, Dose 1 | 54 | 41 | 45 | 54
  Related Irritability, Dose 1: number analyzed (Participants) | 518 | 523 | 508 | 517
  Related Irritability, Dose 1 | 199 | 206 | 213 | 235
  Any Loss of appetite, Dose 1: number analyzed (Participants) | 518 | 523 | 508 | 517
  Any Loss of appetite, Dose 1 | 188 | 208 | 196 | 219
  Grade 3 Loss of appetite, Dose 1: number analyzed (Participants) | 518 | 523 | 508 | 517
  Grade 3 Loss of appetite, Dose 1 | 12 | 11 | 9 | 8
  Related Loss of appetite, Dose 1: number analyzed (Participants) | 518 | 523 | 508 | 517
  Related Loss of appetite, Dose 1 | 95 | 106 | 111 | 117
  Any Temperature, Dose 1: number analyzed (Participants) | 518 | 523 | 508 | 517
  Any Temperature, Dose 1 | 166 | 162 | 170 | 183
  Grade 3 Temperature, Dose 1: number analyzed (Participants) | 518 | 523 | 508 | 517
  Grade 3 Temperature, Dose 1 | 0 | 0 | 0 | 0
  Related Temperature, Dose 1: number analyzed (Participants) | 518 | 523 | 508 | 517
  Related Temperature, Dose 1 | 128 | 119 | 122 | 144
  Any Drowsiness, Dose 2: number analyzed (Participants) | 511 | 515 | 509 | 512
  Any Drowsiness, Dose 2 | 232 | 210 | 231 | 211
  Grade 3 Drowsiness, Dose 2: number analyzed (Participants) | 511 | 515 | 509 | 512
  Grade 3 Drowsiness, Dose 2 | 20 | 20 | 17 | 12
  Related Drowsiness, Dose 2: number analyzed (Participants) | 511 | 515 | 509 | 512
  Related Drowsiness, Dose 2 | 133 | 123 | 137 | 132
  Any Irritability, Dose 2: number analyzed (Participants) | 511 | 515 | 509 | 512
  Any Irritability, Dose 2 | 328 | 312 | 319 | 320
  Grade 3 Irritability, Dose 2: number analyzed (Participants) | 511 | 515 | 509 | 512
  Grade 3 Irritability, Dose 2 | 52 | 35 | 44 | 48
  Related Irritability, Dose 2: number analyzed (Participants) | 511 | 515 | 509 | 512
  Related Irritability, Dose 2 | 208 | 198 | 194 | 212
  Any Loss of appetite, Dose 2: number analyzed (Participants) | 511 | 515 | 509 | 512
  Any Loss of appetite, Dose 2 | 164 | 185 | 183 | 179
  Grade 3 Loss of appetite, Dose 2: number analyzed (Participants) | 511 | 515 | 509 | 512
  Grade 3 Loss of appetite, Dose 2 | 10 | 6 | 6 | 7
  Related Loss of appetite, Dose 2: number analyzed (Participants) | 511 | 515 | 509 | 512
  Related Loss of appetite, Dose 2 | 95 | 103 | 93 | 106
  Any Temperature, Dose 2: number analyzed (Participants) | 511 | 515 | 509 | 512
  Any Temperature, Dose 2 | 146 | 145 | 158 | 144
  Grade 3 Temperature, Dose 2: number analyzed (Participants) | 511 | 515 | 509 | 512
  Grade 3 Temperature, Dose 2 | 1 | 0 | 1 | 1
  Related Temperature, Dose 2: number analyzed (Participants) | 511 | 515 | 509 | 512
  Related Temperature, Dose 2 | 107 | 105 | 116 | 110
  Any Drowsiness, Dose 3: number analyzed (Participants) | 505 | 516 | 505 | 507
  Any Drowsiness, Dose 3 | 181 | 194 | 197 | 193
  Grade 3 Drowsiness, Dose 3: number analyzed (Participants) | 505 | 516 | 505 | 507
  Grade 3 Drowsiness, Dose 3 | 21 | 7 | 13 | 14
  Related Drowsiness, Dose 3: number analyzed (Participants) | 505 | 516 | 505 | 507
  Related Drowsiness, Dose 3 | 112 | 115 | 109 | 112
  Any Irritability, Dose 3: number analyzed (Participants) | 505 | 516 | 505 | 507
  Any Irritability, Dose 3 | 259 | 279 | 271 | 262
  Grade 3 Irritability, Dose 3: number analyzed (Participants) | 505 | 516 | 505 | 507
  Grade 3 Irritability, Dose 3 | 37 | 30 | 32 | 39
  Related Irritability, Dose 3: number analyzed (Participants) | 505 | 516 | 505 | 507
  Related Irritability, Dose 3 | 165 | 178 | 164 | 174
  Any Loss of appetite, Dose 3: number analyzed (Participants) | 505 | 516 | 505 | 507
  Any Loss of appetite, Dose 3 | 149 | 176 | 159 | 154
  Grade 3 Loss of appetite, Dose 3: number analyzed (Participants) | 505 | 516 | 505 | 507
  Grade 3 Loss of appetite, Dose 3 | 14 | 11 | 10 | 9
  Related Loss of appetite, Dose 3: number analyzed (Participants) | 505 | 516 | 505 | 507
  Related Loss of appetite, Dose 3 | 88 | 94 | 83 | 90
  Any Temperature, Dose 3: number analyzed (Participants) | 505 | 516 | 505 | 507
  Any Temperature, Dose 3 | 106 | 127 | 112 | 114
  Grade 3 Temperature, Dose 3: number analyzed (Participants) | 505 | 516 | 505 | 507
  Grade 3 Temperature, Dose 3 | 0 | 2 | 2 | 1
  Related Temperature, Dose 3: number analyzed (Participants) | 505 | 516 | 505 | 507
  Related Temperature, Dose 3 | 71 | 88 | 79 | 89
  Any Drowsiness, Across doses | 376 | 365 | 370 | 377
  Grade 3 Drowsiness, Across doses | 45 | 41 | 40 | 47
  Related Drowsiness, Across doses | 235 | 231 | 235 | 237
  Any Irritability, Across doses | 419 | 436 | 439 | 441
  Grade 3 Irritability, Across doses | 109 | 83 | 86 | 104
  Related Irritability, Across doses | 302 | 304 | 311 | 325
  Any Loss of appetite, Across doses | 295 | 325 | 307 | 312
  Grade 3 Loss of appetite, Across doses | 28 | 23 | 22 | 22
  Related Loss of appetite, Across doses | 180 | 194 | 186 | 182
  Any Temperature, Across doses | 272 | 274 | 277 | 275
  Grade 3 Temperature, Across doses | 1 | 2 | 3 | 2
  Related Temperature, Across doses | 203 | 208 | 208 | 220

44. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms
Description: Assessed solicited general symptoms were drowsiness, irritability, loss of appetite and temperature [defined as rectal temperature greater than or equal to (≥) 38 degrees Celsius (°C)]. Any = occurrence of any general symptoms, regardless of their intensity grade or relationship to study vaccination. Grade 3 Drowsiness = Drowsiness that prevented normal activity. Grade 3 Irritability = Crying that could not be comforted/prevented normal activity. Grade 3 Loss of appetite = Not eating at all. Grade 3 Temperature= temperature above 40.0 (°C). Related = symptom assessed by the investigator as related to the vaccination.
Time Frame: During the 8-day (Days 0-7) post-booster vaccination period
Population: as for outcome 39
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix 3 Group | Nimenrix 2 Group | Menjugate Group | NeisVac-C Group
Number analyzed (Participants) | 491 | 510 | 496 | 504
Participants
  Any Drowsiness | 198 | 206 | 208 | 202
  Grade 3 Drowsiness | 14 | 13 | 21 | 18
  Related Drowsiness | 125 | 129 | 119 | 125
  Any Irritability | 284 | 296 | 284 | 297
  Grade 3 Irritability | 41 | 37 | 37 | 45
  Related Irritability | 180 | 197 | 181 | 186
  Any Loss of appetite | 189 | 193 | 198 | 195
  Grade 3 Loss of appetite | 12 | 21 | 23 | 27
  Related Loss of appetite | 118 | 114 | 114 | 121
  Any Temperature (Rectally) | 187 | 180 | 186 | 170
  Grade 3 Temperature (Rectally) | 2 | 2 | 3 | 7
  Related Temperature (Rectally) | 133 | 132 | 122 | 125

45. Secondary Outcome: Number of Subjects With Any Unsolicited Adverse Events (AEs)
Description: as for outcome 41
Time Frame: Within 31-days (Days 0-30) post-booster vaccination period
Population: as for outcome 39
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix 3 Group | Nimenrix 2 Group | Menjugate Group | NeisVac-C Group
Number analyzed (Participants) | 497 | 511 | 503 | 506
Participants | 179 | 185 | 164 | 167

46. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: Throughout the entire study (from Day 0 to Month 16)
Population: as for outcome 41
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix 3 Group | Nimenrix 2 Group | Menjugate Group | NeisVac-C Group
Number analyzed (Participants) | 528 | 524 | 516 | 527
Participants
  From Day 0 up to Month 1 post-primary vaccination | 1 | 0 | 0 | 0
  From primary vaccination up to ESFU contact | 54 | 56 | 45 | 52

47. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: as for outcome 46
Time Frame: From Booster vaccination (Month 10) up to Extended Safety Follow-Up (ESFU) (Month 16)
Population: as for outcome 39
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix 3 Group | Nimenrix 2 Group | Menjugate Group | NeisVac-C Group
Number analyzed (Participants) | 497 | 511 | 503 | 506
Participants | 14 | 18 | 14 | 17

48. Secondary Outcome: Number of Subjects With New Onset of Chronic Illnesses (NOCIs)
Description: NOCIs assessed included asthma, autoimmune disorders, type 1 diabetes and allergies.
Time Frame: During 31-days (Days 0-30) post-each primary vaccination dose (Day 0 to Month 3) and from primary vaccination up to ESFU (Month 16)
Population: as for outcome 41
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix 3 Group | Nimenrix 2 Group | Menjugate Group | NeisVac-C Group
Number analyzed (Participants) | 528 | 524 | 516 | 527
Participants
  Day 0 - Day 30 after each primary dose | 11 | 6 | 5 | 5
  From primary vaccination up to ESFU contact | 14 | 11 | 15 | 11

49. Secondary Outcome: Number of Subjects With New Onset of Chronic Illnesses (NOCIs)
Description: NOCIs assessed included asthma, autoimmune disorders, type 1 diabetes and allergies.
Time Frame: From Booster vaccination (Month 10 to Month 11) up to ESFU (Month 16)
Population: as for outcome 39
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix 3 Group | Nimenrix 2 Group | Menjugate Group | NeisVac-C Group
Number analyzed (Participants) | 497 | 511 | 503 | 506
Participants | 2 | 2 | 5 | 3

ADVERSE EVENTS:
Time Frame: Solicited local and general symptoms: during the 8-day (Days 0-7) period after each vaccination. Unsolicited adverse events (AEs): during the 31-day (Days 0-30) period after each vaccination. SAEs: throughout the entire study (Day 0-Extended Safety Follow-up at Month 16).
Arm/Group | Nimenrix 3 Group | Nimenrix 2 Group | Menjugate Group | NeisVac-C Group
All-Cause Mortality (participants affected / at risk) | 0/528 | 0/524 | 0/516 | 0/527
Serious Adverse Events (participants affected / at risk) | 54/528 | 56/524 | 45/516 | 52/527
Other Adverse Events (participants affected / at risk) | 512/528 | 516/524 | 506/516 | 513/527
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nimenrix 3 Group (N=528) | Nimenrix 2 Group (N=524) | Menjugate Group (N=516) | NeisVac-C Group (N=527)
Lymphadenitis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Wolff-parkinson-white syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Laryngomalacia (Congenital, familial and genetic disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Plagiocephaly (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis allergic (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aphthous ulcer (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Enteritis (Gastrointestinal disorders) | 0 (0) | 3 (3) | 1 (1) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Inguinal hernia, obstructive (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 5 (5) | 0 (0) | 3 (3)
Milk allergy (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Adenovirus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anal abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atypical pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bacterial pyelonephritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Bronchiolitis (Infections and infestations) | 12 (12) | 10 (10) | 9 (9) | 14 (14)
Bronchitis (Infections and infestations) | 9 (11) | 4 (4) | 1 (1) | 8 (9)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Conjunctivitis bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Croup infectious (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Encephalitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Epstein-barr virus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Exanthema subitum (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 6 (6) | 3 (3) | 5 (5) | 3 (3)
Gastroenteritis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis norovirus (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis rotavirus (Infections and infestations) | 2 (2) | 2 (2) | 1 (1) | 2 (2)
Gastroenteritis salmonella (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Genital candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
H1n1 influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hand-foot-and-mouth disease (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Herpes simplex (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Intervertebral discitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Laryngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Oral candidiasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Otitis media (Infections and infestations) | 3 (3) | 0 (0) | 2 (2) | 1 (1)
Otitis media acute (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 2 (3)
Pertussis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 4 (4) | 3 (3) | 6 (6) | 5 (5)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia respiratory syncytial viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1) | 1 (2) | 1 (2) | 4 (4)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 2 (2) | 3 (3) | 2 (2) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rotavirus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 4 (4) | 2 (2) | 2 (2) | 1 (1)
Urinary tract infection (Infections and infestations) | 3 (3) | 1 (1) | 0 (0) | 2 (2)
Viral infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Viral rash (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 4 (4) | 2 (2)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Near drowning (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skull fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Sacroiliitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Torticollis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebral haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Brain injury (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0) | 1 (2) | 1 (1)
Febrile convulsion (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Hypotonia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Breath holding (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Balanoposthitis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Testicular retraction (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Apparent life threatening event (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Kawasaki's disease (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nimenrix 3 Group (N=528) | Nimenrix 2 Group (N=524) | Menjugate Group (N=516) | NeisVac-C Group (N=527)
Bronchiolitis (Infections and infestations) | 34 (39) | 29 (32) | 31 (33) | 37 (43)
Bronchitis (Infections and infestations) | 45 (49) | 31 (35) | 34 (37) | 48 (56)
Conjunctivitis (Infections and infestations) | 27 (28) | 21 (24) | 31 (32) | 31 (34)
Decreased appetite (Metabolism and nutrition disorders) | 361 (692) | 367 (762) | 355 (738) | 370 (747)
Diarrhoea (Gastrointestinal disorders) | 34 (37) | 31 (39) | 32 (42) | 32 (35)
Erythema (Skin and subcutaneous tissue disorders) | 411 (1036) | 412 (1079) | 432 (1139) | 412 (1100)
Gastroenteritis (Infections and infestations) | 31 (32) | 31 (32) | 21 (22) | 18 (18)
Irritability (Psychiatric disorders) | 446 (1205) | 457 (1230) | 455 (1238) | 460 (1247)
Nasopharyngitis (Infections and infestations) | 25 (30) | 28 (30) | 33 (42) | 30 (35)
Pain (General disorders) | 386 (895) | 379 (899) | 394 (927) | 379 (892)
Pyrexia (General disorders) | 348 (627) | 348 (647) | 349 (660) | 343 (645)
Rhinitis (Infections and infestations) | 33 (39) | 31 (34) | 40 (41) | 21 (24)
Somnolence (Nervous system disorders) | 398 (909) | 386 (892) | 399 (921) | 408 (903)
Swelling (General disorders) | 376 (858) | 380 (864) | 391 (924) | 372 (890)
Upper respiratory tract infection (Infections and infestations) | 108 (146) | 118 (166) | 108 (162) | 103 (135)
Vomiting (Gastrointestinal disorders) | 24 (27) | 20 (22) | 26 (28) | 13 (15)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.